# STATISTICAL ANALYSIS PLAN

VERSION: 1.0 DATE: 12 JANUARY 2021

## **STUDY DRUG:**

DEFIBROTIDE (DEFIBROTIDE SODIUM)

### PROTOCOL/STUDY NUMBER:

JZP395-201 Protocol (09 February 2019)

# **STUDY TITLE:**

Prospective, Multicenter, Open-Label, Single Arm, Phase 2 Study to Evaluate the Safety and Efficacy of Defibrotide in the Prevention of Chimeric Antigen Receptor-T-cell-associated Neurotoxicity in Subjects with Relapsed or Refractory Diffuse Large B-cell Lymphoma Receiving Axicabtagene Ciloleucel (Yescarta®)

#### **SPONSOR:**

Jazz Pharmaceuticals
3170 Porter Dr., Palo Alto, CA 94304

This study is being conducted in compliance with good clinical practice, including the archiving of essential documents.

# SIGNATURE PAGE

This document has been prepared by:

Pl

Jazz Pharmaceuticals

Pl

21-Jan-2021

Date

21-Jan-2021

Date

21-Jan-2021

Date

21-Jan-2021

Date

Jazz Pharmaceuticals

# TABLE OF CONTENTS

| TABLE ( | OF CONTENTS | 3 |
|---|---|---|
| 1. | LIST OF ABBREVIATIONS | 8 |
| 2. | MODIFICATION HISTORY | 9 |
| 3. | INTRODUCTION | 10 |
| 4. | STUDY OBJECTIVES AND ENDPOINTS | 11 |
| 4.1. | Study Objectives | 11 |
| 4.1.1. | Primary Objective | 11 |
| 4.1.2. | Secondary Objectives | 11 |
| 4.1.3. | Exploratory Objectives | 11 |
| 4.2. | Study Endpoints | 11 |
| 4.2.1. | Primary Endpoints | 11 |
| 4.2.2. | Secondary Endpoints | 11 |
| 4.2.3. | Exploratory Endpoints | 12 |
| 5. | STUDY DESIGN | 13 |
| 5.1. | Summary of Study Design | 13 |
| 5.2. | Study Treatment | 14 |
| 5.3. | Power and Sample Size Considerations | 15 |
| 5.4. | Randomization and Blinding | 16 |
| 5.5. | Interim Analysis | 16 |
| 6. | ANALYSIS SETS | 17 |
| 7. | GENERAL ASPECTS FOR STATISTICAL ANALYSIS | 18 |
| 7.1. | General Methods | 18 |
| 7.2. | Baseline and Study Day Definitions | 18 |
| 7.2.1. | Baseline | 18 |
| 7.2.2. | Study Day | 18 |
| 7.2.3. | Visit Windows | 18 |
| 7.2.3.1. | Neurotoxicity Evaluation and CRS Grading at the Primary Efficacy Evaluation Visit | 18 |
| 7.2.3.2. | Adverse Events | 19 |
| 7.2.4. | Missing Data | 19 |
| 7.2.4.1. | Incomplete and Missing AE Start Date | 19 |
| 7.2.4.2. | Incomplete and Missing Prior and Concomitant Medication Start Date | 20 |

| 7.2.4.3. | Incomplete and Missing Prior and Concomitant Medication End Date | 20 |
|---|---|---|
| 7.2.4.4. | Missing Treatment Relationship for AEs and SAEs | 20 |
| 7.2.4.5. | Missing Lymphoma Response | 20 |
| 7.3. | Hypotheses Testing | 20 |
| 7.4. | Level of Significance & Multiplicity Adjustment | 21 |
| 7.5. | Subgroups and Subgroup Analyses | 21 |
| 7.6. | Changes to Planned Analyses | 21 |
| 8. | STUDY POPULATION SUMMARIES | |
| 8.1. | Analysis Sets | 22 |
| 8.2. | Disposition | 22 |
| 8.2.1. | Subject Disposition | 22 |
| 8.2.2. | Defibrotide Disposition | 23 |
| 8.3. | Demographic and Baseline Disease Characteristics | 23 |
| 8.4. | Medical History | 24 |
| 8.5. | Yescarta Administration | 24 |
| 8.6. | Prior and Concomitant Medications | 25 |
| 8.6.1. | Prior Medications | 26 |
| 8.6.2. | Concomitant Medications | 26 |
| 8.6.2.1. | Lymphodepletion Chemotherapy | 26 |
| 8.6.2.2. | Other Concomitant Medications | 27 |
| 8.7. | Protocol Deviations | 27 |
| 9. | EFFICACY | 28 |
| 9.1. | Primary Efficacy Endpoint and Analysis | 28 |
| 9.1.1. | Primary Efficacy Endpoint | 28 |
| 9.1.2. | CTCAE v5.0 Grading of Neurotoxicity | 28 |
| 9.1.3. | Analysis of the Primary Efficacy Endpoint | |
| 9.1.4. | Sensitivity Analyses | 30 |
| 9.1.4.1. | Sensitivity Analysis: Analysis of CAR-T-associated Neurotoxicity of Any Grade Defined by CTCAE v5.0 by CAR-T Day +30 for All Enrolled Subjects Treated at RP2D and Having Yescarta Infusion | 30 |
| 9.1.4.2. | Sensitivity Analysis: Analysis of CAR-T-associated Neurotoxicity of Any Grade Defined by CTCAE v5.0 by CAR-T Day +30 for All Subjects Enrolled at RP2D and Having Yescarta Infusion | 30 |
| 9.1.5. | Subgroup Analyses | |

| 9.2. | Secondary Endpoints and Analyses | 21 |
|---|---|---|
| 9.2.1. | | |
| | Secondary Efficacy Endpoint | 31 |
| 9.2.1.1. | Incidence of CAR-T-associated Neurotoxicity of Grade 3 or Greater Defined by CTCAE v5.0 by CAR-T Day +30 | 31 |
| 9.2.1.2. | Incidence of CAR-T-associated Neurotoxicity (Any Grade and Grade 3 or Greater) according to the ASBMT Consensus Grading System by CAR-T Day +30 | 31 |
| 9.2.1.3. | Incidence of CRS (Any Grade according to the ASBMT Consensus Grading System) by CAR-T Day +30 | 32 |
| 9.2.1.4. | Use of High Dose Steroid by CAR-T Day +30 | 32 |
| 9.2.2. | Sensitivity Analyses | 33 |
| 9.2.3. | Subgroup Analyses | 33 |
| 9.3. | Exploratory Endpoints | 33 |
| 9.3.1. | Duration of Hospital Stay and ICU Stay | 33 |
| 9.3.2. | Duration of CAR-T-associated Neurotoxicity by CTCAE v5.0 | 35 |
| 10. | SAFETY | 36 |
| 10.1. | Exposure | 36 |
| 10.1.1. | Extent of Exposure | 36 |
| 10.1.2. | Treatment Compliance | 37 |
| 10.2. | Adverse Events | 37 |
| 10.2.1. | Dose-limiting Toxicities | 37 |
| 10.2.2. | Adverse Events | 38 |
| 10.2.3. | Adverse Events of Special Interest | 39 |
| 10.2.4. | Adverse Event Summary for Public Disclosure | 39 |
| 10.2.5. | Summary of Adverse Events | 39 |
| 10.3. | Laboratory Assessments | 39 |
| 10.4. | Vital Signs | 40 |
| 10.5. | Lymphoma Response | 41 |
| 11. | PHARMACOKINETIC ANALYSES | 42 |
| 11.1. | General Considerations | 42 |
| 11.2. | Defibrotide Plasma Concentrations | 42 |
| 11.3. | Defibrotide Pharmacokinetic Parameters | 43 |
| 12. | PHARMACODYNAMIC ANALYSES | 46 |
| 13. | COVID-19 | 47 |

# 

# LIST OF TABLES

| Table 1: | List of Abbreviations | 8 |
|----------|-----------------------|---|
|----------|-----------------------|---|

# 1. LIST OF ABBREVIATIONS

Table 1: List of Abbreviations

| Abbreviation | Term |
|--------------|-------------------------------------------------------|
| ASBMT | American Society for Blood and Marrow Transplantation |
| AE | Adverse event |
| ATC | Anatomical therapeutic chemical |
| AUC | Area under the curve |
| AUMC | Area under the first moment curve |
| CAR-T | Chimeric antigen receptor-T-cell |
| CI | Confidence interval |
| CRF | Case report form |
| CRS | Cytokine release syndrome |
| CSR | Clinical study report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DLBCL | Diffuse large B-cell lymphoma |
| DLT | Dose-limiting toxicity |
| HLGT | High Level Group Term |
| ICE | Immune effector cell-associated encephalopathy |
| ICH | International Conference on Harmonisation |
| ICU | Intensive care unit |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MLE | Maximum likelihood estimate |
| PK | Pharmacokinetics |
| PT | Preferred term |
| RP2D | Recommended phase 2 dose |
| SAC | Safety Assessment Committee |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SAS | Statistical Analysis System |
| SMQ | Standardised MedDRA Query |
| SOC | System organ class |

| TEAE | Treatment-emergent adverse event |
|-------|------------------------------------------|
| TESAE | Treatment-emergent serious adverse event |

# 2. MODIFICATION HISTORY

Version History:

| Version Date Description | | Description |
|--------------------------|-----------------|-------------|
| Original | 12 January 2021 | |

#### 3. INTRODUCTION

The purpose of this statistical analysis plan (SAP) is to describe in detail the statistical methodology and planned analyses for Protocol JZP395-201 for inclusion in the clinical study report (CSR). Mock tables, listings, and figure shells will be provided in a separate supporting document.

This SAP complies with the International Conference on Harmonisation (ICH) Harmonised Tripartite Guideline Topic E9, Statistical Principles for Clinical Trials. The current version of the SAP is based on the following study documents:

- Original Protocol, dated 09 February 2019
- Case report form (CRF), Version dated 05 December 2019

Any additional analyses or deviation from the analyses outlined in this plan will be documented with rationale in the final CSR. All decisions regarding the final analysis of the study results, as defined in this SAP, have been made prior to database lock of the study data.

#### 4. STUDY OBJECTIVES AND ENDPOINTS

# 4.1. Study Objectives

# 4.1.1. Primary Objective

The primary objective of the study is to assess the efficacy of defibrotide for the prevention of chimeric antigen receptor-T-cell-associated (CAR-T-associated) neurotoxicity in subjects with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) receiving Yescarta.

## 4.1.2. Secondary Objectives

- To further assess the efficacy of defibrotide for the prevention of CAR-T-associated neurotoxicity in subjects with relapsed or refractory DLBCL receiving Yescarta
- To assess the safety of defibrotide for the prevention of CAR-T-associated neurotoxicity in subjects with relapsed or refractory DLBCL receiving Yescarta
- To assess the pharmacokinetics (PK) of defibrotide

# 4.1.3. Exploratory Objectives

- Biomarker analysis before and after defibrotide
- Biomarker analysis before and after Yescarta
- Duration of hospital stay and intensive care unit (ICU) stay

# 4.2. Study Endpoints

# 4.2.1. Primary Endpoints

The primary endpoint of the study is the incidence of CAR-T-associated neurotoxicity (any grade, defined by Common Terminology Criteria for Adverse Events [CTCAE] v5.0) by CAR-T Day +30.

# 4.2.2. Secondary Endpoints

- The secondary efficacy endpoints of the study are as follows:
  - Incidence of CAR-T-associated neurotoxicity of Grade 3 or greater defined by CTCAE v5.0 by CAR-T Day +30
  - Incidence of CAR-T-associated neurotoxicity (any grade and Grade 3 or greater) according to the ASBMT consensus grading system (Lee et al. 2019) by CAR-T Day +30
  - Incidence of cytokine release syndrome (CRS; any grade, according to the ASBMT consensus grading system [Lee et al. 2019]) by CAR-T Day +30
  - Use of high dose steroid by CAR-T Day +30
- The following safety endpoints will be evaluated as secondary endpoints of the study:
  - Incidence of TEAEs that occur up to 30 days after the last dose of defibrotide

- Incidence of TESAEs that occur up to 30 days after the last dose of defibrotide
- Lymphoma response evaluation by Cheson criteria (Cheson et al. 2016) up to CAR-T Day +60
- PK of defibrotide

# 4.2.3. Exploratory Endpoints

The following exploratory endpoints will be evaluated:

- Biomarker analysis before and after defibrotide
- Biomarker analysis before and after Yescarta
- Duration of hospital stay and ICU stay

#### 5. STUDY DESIGN

# 5.1. Summary of Study Design

This is a prospective, open-label, single-arm study evaluating the safety and efficacy of defibrotide for the prevention of CAR-T-associated neurotoxicity in subjects with relapsed or refractory DLBCL receiving Yescarta. The primary endpoint of the study is the incidence of CAR-T-associated neurotoxicity (any grade, defined by CTCAE v5.0) by CAR-T Day +30.

This is a 2-part study starting with a safety lead-in phase (Part 1) that will determine the recommended phase 2 dose (RP2D) to be used in all subsequent eligible subjects (Part 2). Part 1 of the study is based on a standard 3 + 3 design and will evaluate the safety of a 2.5 mg/kg/dose regimen of defibrotide in 3 to 6 eligible subjects before escalating to a 6.25 mg/kg/dose regimen in 3 to 6 eligible subjects, according to the algorithm shown in Figure 1. A Safety Assessment Committee (SAC) will be formed to determine the dose-limiting toxicities (DLTs) during Part 1 of the study. After the RP2D is established, Part 2 will enroll subjects to obtain a total of approximately 32 subjects treated at the RP2D, including those who were treated at the RP2D in Part 1. It is projected that 10% of enrolled subjects will not receive CAR-T treatment (Yescarta), and therefore, will not contribute to the primary efficacy analysis, ie, 29 of the 32 subjects treated at the RP2D will be efficacy evaluable (see definition of the Efficacy Evaluable Analysis Set in Section 6).

Figure 1: Dose Escalation Algorithm



<sup>\*</sup>Efficacy evaluable; Subjects in Part 1 treated at the RP2D will be included in the efficacy and safety analyses.

An SAC will be formed for determination of any DLTs during Part 1 of the study. The SAC will continue monitoring safety in Part 2 of the study. The SAC will include the Sponsor's Study Medical Monitor, Study Biostatistician, Pharmacovigilance Physician, and Principal Investigators. The Sponsor's Study Medical Monitor will be the chair of the SAC. All roles and responsibilities of the SAC, as well as the timing of safety reviews, will be fully described in a SAC charter.

The significant toxicity from CAR-T treatment may not be distinguishable from TEAEs attributable to defibrotide, as the safety profile of defibrotide in this patient population has not been characterized. During Part 1 of the study, all TEAEs that occur from the start of the first dose of defibrotide up to 7 days after the last dose of defibrotide will be first screened for DLT by the principal investigator of the site where the event occurred and by the Sponsor. The final determination of DLT will then be made by the SAC from TEAEs considered to have a causal relationship to defibrotide. As an exception, all bleeding TEAEs, regardless of relationship to defibrotide, will be evaluated by the SAC as potential DLTs. Because all hemorrhagic events are considered adverse drug reactions of defibrotide, the SAC will focus on any grade of intracranial hemorrhage and any other hemorrhage of Grade 2 or greater, per CTCAE v5.0. Of note, CAR-T-associated neurotoxicity is not a DLT.

The study duration is expected to be approximately 21 months, with an estimated enrollment period of 18 months and participation for each subject of approximately 3 months. Each subject is considered to have completed the study once the CAR-T Day +37 visit is completed and lymphoma response data are available; if lymphoma response data are not available by CAR-T Day +60, the subject is considered to have completed the study on CAR-T Day +60. End of study for each subject is the time at which the subject completes the study, the time of death, lost to follow-up, or early termination from the study. The study is considered completed once all enrolled subjects have reached the end of study. The final analysis to support the CSR will take place after study completion.

# **5.2.** Study Treatment

Subjects will receive defibrotide at 2.5 mg/kg/dose or 6.25 mg/kg/dose, lymphodepletion chemotherapy (per the investigator's standard of care), and Yescarta (per labeled use).

Defibrotide solution is administered intravenously by study site personnel at 2.5 mg/kg/dose or 6.25 mg/kg/dose. Each defibrotide dose should be infused over 2 hours  $\pm$  15 minutes. Individual doses of defibrotide are determined for individual subjects based on body weight at baseline, which in this study is defined as the date of the first defibrotide infusion, prior to initiation of infusion. To facilitate efficient drug administration, each dose will be rounded to the nearest 10 mg for subjects weighing  $\geq$  35 kg and the nearest 5 mg for subjects weighing  $\leq$  35 kg.

To minimize the endothelial damage from lymphodepletion chemotherapy, defibrotide is to start on the first day (CAR-T Day -5 [Study Day 1]; see definition of Study Day in Section 7.2.2) of lymphodepletion chemotherapy (with 1 administration of defibrotide per day) and continue for 3 days (with administration of defibrotide on each day occurring immediately prior to lymphodepletion chemotherapy). The window between the end of defibrotide infusion and start of lymphodepletion chemotherapy should not exceed 2 hours. On CAR-T Day -2 (Study Day 4) and CAR-T Day -1 (Study Day 5), defibrotide will not be administered. Starting on CAR-T Day 0 (Study Day 6), defibrotide will be administered every 6 hours (4 times a day) until CAR-T Day +7 (Study Day 13). A minimum of 2 doses of defibrotide must be administered prior to Yescarta infusion on CAR-T Day 0. Yescarta may be delayed for up to 2 days, in which case CAR-T Day 0 will correspond to Study Day 7 (1-day delay) or Study Day 8 (2-day delay).

Each defibrotide dose (infused over an infusion period of 2 hours  $\pm$  15 minutes) may be administered within  $\pm$  1 hour of the scheduled dosing time, provided that there is at least a 2-hour window between the end of an infusion and the start of the next infusion.

This dosing schedule is summarized in the table below:

#### **Schedule of Defibrotide Dosing**

| | Outpatient | | | Inpatient required | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| CAR-T Day | -5 | -4 | -3 | -2 | -1 | 0<br>(+2 days) <sup>a</sup> | +1 to +7<br>(+2 days) <sup>a</sup> | +8 to +37<br>(+2 days) <sup>a</sup> | +60<br>(+2 days) <sup>a</sup> |
| Study Day | 1 | 2 | 3 | 4 | 5 | 6 | 7-13 | 14-43 | 66 |
| Lymphodepletion chemotherapy | X <sup>b</sup> | X <sup>b</sup> | X <sup>b</sup> | | | | | | |
| Yescarta | | | | | | X <sup>c</sup> | | | |
| Defibrotide <sup>d</sup> | QD <sup>e</sup> | QD <sup>e</sup> | QD <sup>e</sup> | | | QID <sup>f</sup> | QID <sup>f</sup> | | |

Abbreviations: CAR-T = chimeric antigen receptor T-cell; QD = once daily; QID = 4 times a day.

If a subject develops any grade intracranial hemorrhage or any other hemorrhage of Grade 2 or greater, defibrotide must be discontinued. In addition, discontinuation of defibrotide is recommended for subjects that need to undergo surgery or invasive procedures. If a subject experiences Grade 3 or greater CAR-T-associated neurotoxicity, the treatment must discontinue, as such an event is considered failure to prevent CAR-T-associated neurotoxicity. Subjects who discontinue defibrotide due to toxicity must not resume defibrotide treatment on this study but should still continue protocol defined evaluations as long as the subject remains on the study.

# **5.3.** Power and Sample Size Considerations

Part 1 of the study will determine the RP2D by evaluating the safety of defibrotide in subjects receiving CAR-T-cell therapy (Yescarta). Two cohorts (2.5 mg/kg/dose and 6.25 mg/kg/dose) will be evaluated in a standard 3 + 3 design. If DLTs are observed in greater than 1 out of 3 or greater than 1 out of 6 subjects under the same dose level, then the dose is considered not safe. The highest dose that is determined to be safe (ie, the RP2D) will be given to subjects enrolled in Part 2 of the study and will be evaluated for the safety and efficacy of defibrotide for prevention of CAR-T-associated neurotoxicity. Subjects treated at the RP2D in Part 1 will be included in the efficacy and safety analyses of the study.

The primary objective of the study is to assess the efficacy of defibrotide for the prevention of CAR-T-associated neurotoxicity. Simon's optimal 2-stage design (Simon 1989) is employed to test the incidence rate of CAR-T-associated neurotoxicity by CAR-T Day +30 in the target patient population, in order to avoid unnecessarily exposing subjects to a non-efficacious therapy. The historical rate of CAR-T-associated neurotoxicity is 64% (Neelapu et al. 2017); it is hypothesized that administration with defibrotide will reduce this by half, to a CAR-T-associated neurotoxicity

<sup>&</sup>lt;sup>a</sup> Yescarta may be delayed for up to 2 days, in which case CAR-T Day 0 will correspond to Study Day 7 (1-day delay) or Study Day 8 (2-day delay).

<sup>&</sup>lt;sup>b</sup> Per the investigator's standard of care.

<sup>&</sup>lt;sup>c</sup> Per the labeled use.

<sup>&</sup>lt;sup>d</sup> Defibrotide should be administered within ±1 hour of the scheduled dose, provided that there is at least a 2-hour window between the end of an infusion and the start of the next infusion.

<sup>&</sup>lt;sup>e</sup> Defibrotide must be administered immediately prior to lymphodepletion chemotherapy. The window between the end of defibrotide infusion and start of lymphodepletion chemotherapy should not exceed 2 hours.

f At least 2 doses of defibrotide must be administered on CAR-T Day 0 (Study Day 6) prior to administration of Yescarta.

rate of 32% (ie, a no CAR-T-associated neurotoxicity rate of 68%). The sample size calculation is based on testing the null and alternative hypotheses (see details in Section 7.3) with an overall 1-sided Type I error rate of 0.05 and a statistical power of at least 92% when the rate of no CAR-T-associated neurotoxicity rate is  $\geq$  68%. In the first stage, 10 efficacy evaluable subjects will be accrued. If there are 4 or fewer subjects without CAR-T-associated neurotoxicity post-CAR-T-cell therapy in these 10 subjects, the study will be stopped. Otherwise, 19 additional efficacy evaluable subjects will be accrued for a total of 29. The null hypothesis will be rejected if 15 or more subjects without CAR-T-associated neurotoxicity post-CAR-T-cell therapy are observed in these 29 subjects.

The total sample size of the study comprises the sum of subjects from Part 1 of the study, and those from Part 2 of the study. Subjects treated at the RP2D in Part 1 will be included in the efficacy and safety analyses. Under the assumption that defibrotide is safe at one of the 2 dose levels tested, the maximum number of subjects in Part 1 is 12, with 6 treated at the RP2D; the minimum is 9, with 6 treated at the RP2D. Allowing for 10% of enrolled subjects to be non-eligible for the efficacy evaluation (ie, not in the Efficacy Evaluable Analysis Set), a planned maximum total of 38 subjects and a planned minimum total of 35 will be required. Additional subjects may be enrolled to provide 29 efficacy evaluable subjects.

# 5.4. Randomization and Blinding

Randomization is not applicable, as this is a single-arm study.

Blinding is not applicable in this open-label study.

# 5.5. Interim Analysis

No formal interim analysis is planned for this study.

# 6. ANALYSIS SETS

For purposes of analysis, the following populations are defined:

| Analysis Set | Description |
|---|---|
| Enrolled | All subjects who signed the informed consent form and met all eligibility criteria for the study |
| Safety | The Safety Analysis Set will include all enrolled subjects who received at least 1 dose of defibrotide. |
| Enrolled (RP2D) | The Enrolled (RP2D) Analysis Set will include all enrolled subjects treated with at least 1 dose of defibrotide at the RP2D and having Yescarta infusion. |
| Efficacy Evaluable | The Efficacy Evaluable Analysis Set will consist of all subjects in the Enrolled (RP2D) Analysis Set: |
| | <ul> <li>who received at least 18 doses (of all 35) of defibrotide<br/>and either</li> </ul> |
| | <ul> <li>developed CAR-T-associated neurotoxicity on or<br/>before CAR-T Day +30; OR</li> </ul> |
| | - completed the CAR-T Day +30 neurological assessment; |
| | AND |
| | <ul> <li>who discontinued defibrotide due to CAR-T-associated<br/>neurotoxicity before receiving 18 doses of defibrotide.</li> </ul> |
| | In addition, subjects must NOT have their Yescarta infusion delayed by more than 2 days from the original schedule. |
| PK | The PK Analysis Set will include all subjects who received at least 1 dose of defibrotide and had at least 1 evaluable PK concentration. |
| PK Evaluable | The PK Evaluable Analysis Set will include all subjects in the PK Analysis Set whose key PK parameters such as area under the curve (AUC), CL, and $t_{1/2}$ can be determined for the CAR-T Day -5 visit (see Section 11.3 for the definitions of CL and $t_{1/2}$ ). |

#### 7. GENERAL ASPECTS FOR STATISTICAL ANALYSIS

The statistical principles applied in the design and planned analyses of this study are consistent with ICH E9 guidelines (ICH 1998).

#### 7.1. General Methods

All study data will be summarized using descriptive statistics (sample size, mean, standard deviation, median, minimum, and maximum) for continuous variables (eg, age, weight) and using the number and percentage of subjects for categorical variables (eg, sex, race), unless otherwise specified. Data listings will be organized by study part (by cohort within Part 1) and then by subject within each cohort in Part 1 and Part 2.

All summaries, statistical analyses, and data listings described below will be completed using Version 9.4 or later of the Statistical Analysis System (SAS Institute, Inc., Cary, NC).

# 7.2. Baseline and Study Day Definitions

#### 7.2.1. Baseline

For procedures and assessments, baseline is defined as the date of the first defibrotide infusion (ie, Study Day 1 or CAR-T Day -5 as defined in Section 7.2.2), prior to initiation of infusion.

For safety analyses, baseline is defined as the same as above.

For efficacy analyses, baseline is defined as the date of CAR-T-cell therapy (Yescarta) infusion (ie, CAR-T Day 0 as defined in Section 7.2.2).

# **7.2.2. Study Day**

Study Day 1 is defined as the date of the first defibrotide infusion. For this study, the schedule of procedures and assessments will also reference the day relative to CAR-T Day 0, which is defined as the date of CAR-T-cell therapy (Yescarta) infusion. For example, Study Day 1 of this study will also be referred to as CAR-T Day -5, whereas the date of Yescarta infusion, CAR-T Day 0 will also be referred to as Study Day 6. Yescarta infusion may be delayed for up to 2 days, in which case CAR-T Day 0 will correspond to Study Day 7 (1-day delay) or Study Day 8 (2-day delay). Refer to the defibrotide dosing schedule table in Section 5.2.

#### 7.2.3. Visit Windows

# 7.2.3.1. Neurotoxicity Evaluation and CRS Grading at the Primary Efficacy Evaluation Visit

For the neurotoxicity evaluation and CRS grading at the primary efficacy evaluation visit scheduled on CAR-T Day +30, an analysis window of + 3 days will be used to identify the last assessments to be used for the analyses of the secondary efficacy endpoints according to the ASBMT consensus grading system. The upper limit of the analysis window is CAR-T Day +33. All valid non-missing assessments from CAR-T Day 0 up to CAR-T Day +33 will be used in the analyses.

#### 7.2.3.2. Adverse Events

For the adverse event (AE) evaluations at the primary efficacy evaluation visit scheduled on CAR-T Day +30 and at the final safety follow-up visit scheduled on CAR-T Day +37, the table below provides the upper limits of the analysis windows for the purpose of identifying the last assessments to be used in the analyses.

| Visit Identifier | Upper Limit |
|------------------|---------------|
| CAR-T Day +30 | CAR-T Day +33 |
| CAR-T Day +37 | CAR-T Day +43 |

All valid non-missing assessments from CAR-T Day 0 to CAR-T Day +33 will be used for the analyses of the primary and secondary efficacy endpoints based on CTCAE v5. All valid non-missing assessments from the date of the first defibrotide infusion to CAR-T Day +43 will be used for the safety analyses.

# 7.2.4. Missing Data

Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument. These data will be indicated by the use of a "blank" in subject listing displays. Note that if any missing data is imputed, the imputed data will only be used in summaries, and will not be included in any listing. Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should not be displayed as missing.

#### 7.2.4.1. Incomplete and Missing AE Start Date

For this study, the first dose date is defined the same as baseline for the safety analysis (ie, the date of the first defibrotide infusion). The following imputation rules will be followed, when the AE start date is incomplete (eg, only *year* is present, but *month* and *day* are missing) or completely missing:

- If year is missing (including the situation where the start date is completely missing), set the date to the first dose date.
- If year is present, and month and day are missing, or year and day are present, and month is missing,
  - if *year* = year of first dose, set the date to the first dose date;
  - if year < year of first dose, set month and day to December 31;
  - if *year* > year of first dose, set *month* and *day* to January 1.
- If year and month are present, and day is missing,
  - if year = year of first dose, and
    - if month = month of first dose, set day to day of first dose;
    - if month < month of first dose, set day to the last day of month;
    - if month > month of first dose, set day to the first day of month;

- if *year* < year of first dose, set *day* to the last day of *month*;
- if *year* > year of first dose, set *day* to the first day of *month*.

For all other cases that are not covered above, set the date to the first dose date.

# 7.2.4.2. Incomplete and Missing Prior and Concomitant Medication Start Date

The following imputation rules will be followed, when the prior and concomitant medication start date is incomplete (eg, only *year* is present, but *month* and *day* are missing) or completely missing:

- If year is missing (including the situation where the start date is completely missing), do not impute, and the start date will be treated as missing in the analysis.
- If year is present, and month and day are missing, or year and day are present, and month is missing, set month and day to January 1.
- If year and month are present, and day is missing, set day to the first day of month.

## 7.2.4.3. Incomplete and Missing Prior and Concomitant Medication End Date

The following imputation rules will be followed, when the prior and concomitant medication end date is incomplete (eg, only *year* is present, but *month* and *day* are missing) or completely missing:

- If it is indicated that the concomitant medication is ongoing (ie, "Yes" is checked for the question "Ongoing?" in the CRF), do not impute, since there should not be an end date for this concomitant medication.
- If year is missing (including the situation where the end date is completely missing), do not impute, and the end date will be treated as missing in the analysis.
- If year is present, and month and day are missing, or year and day are present, and month is missing, set month and day to December 31.
- If year and month are present, and day is missing, set day to the last day of month.

## 7.2.4.4. Missing Treatment Relationship for AEs and SAEs

Subjects with the designation of treatment relationship for AEs and SAEs missing will have the worst case scenario assumed to impute the relationship. For subjects who receive defibrotide, if relationship to the study drug (defibrotide) is missing, the event will be assumed to be related to defibrotide.

#### 7.2.4.5. Missing Lymphoma Response

For the analysis of lymphoma response up to CAR-T Day +60, missing data on lymphoma response will be handled using a "Missing = Failure" approach.

# 7.3. Hypotheses Testing

The primary endpoint of the study will be evaluated by the proportion of the study subjects treated at the RP2D who did not develop any CAR-T-associated neurotoxicity by CAR-T Day +30 using the Efficacy Evaluable Analysis Set. The rate of no CAR-T-associated neurotoxicity, denoted by p, will be tested against a pre-defined threshold, 36%, using the rejection rule based on Simon's optimal 2-stage design.

```
Jazz Pharmaceuticals
{Statistical Analysis Plan - Protocol #}
```

Symbolically, this is expressed as follows,

```
H<sub>0</sub>: p \le 36\% (ie, the rate of CAR-T-associated neurotoxicity is more than 64%) versus
```

 $H_a$ : p > 68% (ie, the rate of CAR-T-associated neurotoxicity is no more than 32%).

The null hypothesis will be tested using a 1-sided test with a Type I error rate of 0.05.

# 7.4. Level of Significance & Multiplicity Adjustment

The Type I error rate for testing the null hypothesis for the analysis of the primary endpoint is 0.05, 1-sided (Section 7.3). There will be no adjustments for multiple testing in the analyses for this study.

# 7.5. Subgroups and Subgroup Analyses

Not applicable.

# 7.6. Changes to Planned Analyses

Study objectives are not clearly defined in the protocol. Study objectives are defined in this document corresponding to the study endpoints (see Sections 4.1 and 4.2).

In the protocol, the All Enrolled Analysis Set is defined as all enrolled subjects treated at the RP2D. In this document, this analysis set is renamed and redefined for clarity as the following: The Enrolled (RP2D) Analysis Set is defined as all enrolled subjects treated at the RP2D with at least 1 dose of defibrotide and having Yescarta infusion (see Section 6). Two sensitivity analyses are defined, with one based on the Enrolled (RP2D) Analysis Set and the other based on all subjects enrolled at RP2D and having Yescarta infusion. The latter includes all subjects in the Enrolled (RP2D) Analysis Set and subjects who did not receive any defibrotide.

As the study goes on, the duration of CAR-T-associated neurotoxicity has been identified as of clinical importance. The following analyses have been added accordingly (see Section 9.3.2):

- Analysis of Duration of CAR-T-associated Neurotoxicity of Any Grade Defined by CTCAE v5.0 for All Efficacy Evaluable Subjects
- Analysis of Duration of CAR-T-associated Neurotoxicity of Grade or Greater Defined by CTCAE v5.0 for All Efficacy Evaluable Subjects

#### 8. STUDY POPULATION SUMMARIES

Summaries will be produced by dose level for Part 1, for the phase 2 part of the study and overall, using the Safety Analysis Set unless otherwise specified. For Part 1, there will be no statistical comparison between the 2 dose levels for any of the measures in this section. For the phase 2 part, summaries will be provided for all subjects treated at the RP2D. Note that since subjects treated at the RP2D in Part 1 will also be included in the phase 2 part under the 2-stage design, those subjects will be included in the summaries for both Part 1 and the phase 2 part.

# 8.1. Analysis Sets

All analysis sets will be summarized. The Enrolled Analysis Set will be summarized overall only. The Enrolled (RP2D) and Efficacy Evaluable Analysis Sets will be summarized for the phase 2 part and overall only. The number of subjects screened and enrolled by center and reasons for screen failures will be summarized separately overall only. The following summaries will be provided:

- Analysis Sets by Study Phase and Overall
- Screened and Enrolled Subjects by Center
- Reasons for Screen Failures

Additionally, summaries for public disclosure will tabulate subjects enrolled by country and site and by age category using the Enrolled Analysis Set. The following summaries will be provided:

- Number of Subjects Enrolled by Country and Site
- Number of Subjects Enrolled by Age Category

The following listing will be provided:

• Reasons for Screen Failures

# 8.2. Disposition

#### 8.2.1. Subject Disposition

A summary of subject disposition, including study completion, study withdrawal, and primary reason for study withdrawal, will be provided:

• Subject Disposition by Study Phase and Overall

Every category will be kept in the summary even if it has 0 subjects. Additionally, a disposition summary will be provided using the Enrolled Analysis Set:

• Study Disposition (for Public Disclosure)

The following listing of subject disposition will be provided with date of screening/Study Day, date of enrollment/Study Day, study part, study completion (Yes or No), the last on-study date/Study Day/CAR-T Day and primary reason for study withdrawal (if No to study completion):

• Subject Disposition

If a subject completes the study per protocol, the last on-study date is the last visit date for this subject; if a subject terminates the study early, the date entered in the early termination folder in EDC is the last on-study date for this subject.

## 8.2.2. Defibrotide Disposition

A summary of defibrotide disposition, including defibrotide completion, defibrotide premature discontinuation, and primary reason for defibrotide premature discontinuation, will be provided:

• Defibrotide Disposition by Study Phase and Overall

Every category will be kept in the summary even if it has 0 subjects. The following listing of defibrotide disposition will be provided with the first dose date/Study Day/CAR-T Day, the start date of Yescarta administration/Study Day, the last dose date/Study Day/CAR-T Day, defibrotide completion (Yes or No), and primary reason for defibrotide premature discontinuation (if No to defibrotide completion):

• Defibrotide Disposition

# 8.3. Demographic and Baseline Disease Characteristics

A summary of demographic and baseline disease characteristics will be provided:

• Demographic and Baseline Disease Characteristics by Study Phase and Overall

The following demographic and baseline disease characteristics will be included in the summary:

- o Age in years at baseline (as a continuous variable)
- Age group at baseline (18-64 or  $\ge$  65 years)
- o Sex at birth (Female or Male)
- Race (American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, White, Declined to state, or Mutiple)
- o Ethnicity (Hispanic or Latino, Not Hispanic or Latino, or Declined to state)
- Weight in kg at baseline
- o Eastern Cooperative Oncology Group performance status at baseline (0, 1, 2, 3, or 4)
- Neurotoxicity evaluation at baseline
  - Immune effector cell-associated encephalopathy (ICE) score (Grade 0, Grade 1, Grade 2, Grade 3, or Grade 4)
  - Depressed level of consciousness (Grade 0, Grade 1, Grade 2, Grade 3, or Grade 4)
  - Seizure (Grade 0, Grade 3, or Grade 4)
  - Motor findings (Grade 0, or Grade 4)
  - Raised intracranial pressure/cerebral edema (Grade 0, Grade 3, or Grade 4)
- CRS at baseline
  - Hypotension (Grade 1, Grade 2, Grade 3, or Grade 4)

- Hypoxia (Grade 1, Grade 2, Grade 3, or Grade 4)
- Disease history
  - Time in days between the date of initial diagnosis and baseline
  - Number of previous treatment regimens
  - Primary refractory disease (Yes or No)
  - Refractory to the previous treatment (less than partial response after last treatment; Yes or No)
  - Previous autologous stem cell transplant (Yes or No)
  - Number of recurrences (defined as number of previous treatment regimens 1)

For race, if multiple options are checked, the subject will be categorized under "Multiple". For the ICE score, Grade 0 in a specific category is defined as no toxicity. The following listing of all demographic and baseline disease characteristics specified above will be provided:

• Demographic and Baseline Disease Characteristics

# 8.4. Medical History

Medical history includes diseases and conditions by standard body systems, and information on resolved conditions, intermittent conditions, concurrent illnesses, and previous surgeries. Medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) 21.1. A summary of medical history by system organ class (SOC) and preferred term (PT) will be provided:

Medical History by Study Phase and Overall

System organ classes will be ordered alphabetically, with PTs within an SOC sorted in descending order of incidence in overall. The following listing of medical history will be provided with the start date, ongoing (Yes or No), and the end date, if not ongoing:

Medical History

#### 8.5. Yescarta Administration

Information pertaining to Yescarta administration, including the start date of Yescarta infusion in terms of Study Day (Study Day 6, Study Day 7 or Study Day 8) and infused cell count, will be summarized:

• Yescarta Administration by Study Phase and Overall

The numbers of subjects who did not receive Yescarta and whose Yescarta administration got delayed for more than 2 days will also be included in the summary. Note that for the phase 2 part of the study, subjects who did not receive Yescarta and whose Yescarta administration got delayed for more than 2 days are not efficacy evaluable. The following listing of Yescarta administration will be provided with the start date/Study Day and time, the end date/Study Day and time, and infused cell count (unit):

• Yescarta Administration

#### **8.6.** Prior and Concomitant Medications

Prior medications are defined as all medications and therapies received between the date of the first screening procedure and baseline (but not during treatment with defibrotide), and all prior therapies for the primary disease taken within 90 days prior to signing of the initial informed consent form, inclusive. Concomitant medications are defined as all medications and therapies taken between baseline (for safety analyses) and 30 days after the last dose of defibrotide, inclusive, including lymphodepletion chemotherapy, and medications and therapies started before treatment with defibrotide and continuing on or after the first dose of defibrotide. For reporting purpose, the following approach will be used to determine prior or concomitant medications, after the imputation rules for all incomplete and missing start and end dates (Sections 7.2.4.2 and 7.2.4.3) are applied:

| Start Date | End Date | Decision |
|---|---|---|
| Before baseline | Before baseline | Prior medication |
| Missing | Before baseline | Prior medication |
| Before baseline | On or after baseline | Prior and concomitant medication |
| Baseline to 30 days after the last dose of defibrotide | On or after baseline | Concomitant medication |
| Baseline to 30 days after the last dose of defibrotide | Missing | Concomitant medication |
| Before baseline | Missing, but Ongoing = No at or before baseline | Prior medication |
| Before baseline | Missing, but Ongoing = No after baseline | Prior and concomitant medication |
| Before baseline | Missing, but Ongoing = Yes | Prior and concomitant medication |
| Before baseline | Missing, and Ongoing (Yes or No) not answered | Prior and concomitant medication |
| Missing | On or after baseline | Prior and concomitant medication |
| Missing | Missing, but Ongoing = No at or before baseline | Prior medication |
| Missing | Missing, but Ongoing = No after baseline | Prior and concomitant medication |
| Missing | Missing, but Ongoing = Yes | Prior and concomitant medication |

| Missing | Missing, and Ongoing (Yes or No) not answered | Prior and concomitant medication |
|---|---|---|
| | ′ | |

Prior and concomitant medications will be coded using the World Health Organization drug dictionary (WHODRUG C3 Global 2019Q1), and summarized separately by the generic name. Medications that are not coded will only be listed.

#### **8.6.1.** Prior Medications

Information regarding prior medications is collected on the Prior and Concomitant Medications page of the CRF. A summary of prior medications will be provided:

Prior Medications by Study Phase and Overall

The summary of prior medications will be provided by anatomical therapeutic chemical (ATC) 4<sup>th</sup> level and PT, and ATCs will be ordered alphabetically, with PTs within an ATC sorted in descending order of incidence in overall. Subjects reporting more than 1 prior medication will be counted only once in the total number of subjects taking a prior medication. Prior medications will be sorted in descending order of incidence in overall. The following listing of prior medications will be provided with ATC 4<sup>th</sup> level classification, PT, indication, the start date, ongoing (Yes or No), the end date, if not ongoing, dose (unit), frequency, and route:

Prior Medications

#### **8.6.2.** Concomitant Medications

Information regarding concomitant medications is collected on the Prior and Concomitant Medications page of the CRF. Concomitant medications will be summarized separately for lymphodepletion chemotherapy (Section 8.6.2.1) and other concomitant medications (Section 8.6.2.2). For each summary, subjects reporting medications with the same generic name 2 or more times will be counted only once for that generic name, and subjects reporting more than 1 concomitant medication will be counted only once in the total number of subjects taking a concomitant medication.

#### **8.6.2.1.** Lymphodepletion Chemotherapy

Lymphodepletion chemotherapy includes cyclophosphamide and fludarabine. A summary of lymphodepletion chemotherapy will be provided:

• Concomitant Medications: Lymphodepletion Chemotherapy by Study Phase and Overall

The summary of lymphodepletion chemotherapy will be provided by ATC 4<sup>th</sup> level and PT, and ATCs will be ordered alphabetically, with PTs within an ATC sorted in descending order of incidence in overall. The following listing of lymphodepletion chemotherapy will be provided with ATC 4<sup>th</sup> level classification, PT, indication, the start date, ongoing (Yes or No), the end date, if not ongoing, dose (unit), frequency, and route:

• Concomitant Medications: Lymphodepletion Chemotherapy

#### **8.6.2.2.** Other Concomitant Medications

Other concomitant medications include concomitant medications other than lymphodepletion chemotherapy. A summary of other concomitant medications will be provided:

• Concomitant Medications: Other (Lymphodepletion Chemotherapy Excluded) by Study Phase and Overall

The summary of other concomitant medications will be provided by ATC 4<sup>th</sup> level and PT, and ATCs will be ordered alphabetically, with PTs within an ATC sorted in descending order of incidence in overall. The following listing of other concomitant medications will be provided with ATC 4<sup>th</sup> level classification, PT, indication, the start date, ongoing (Yes or No), the end date, if not ongoing, dose (unit), frequency, and route:

• Concomitant Medications: Other (Lymphodepletion Chemotherapy Excluded)

## 8.7. Protocol Deviations

Major protocol deviations will be summarized:

• Major Protocol Deviations by Study Phase and Overall

The summary will include but not be limited to the following categories:

- o Inclusion/exclusion criteria
- Informed consent procedure
- Concomitant medication/therapy
- Laboratory assessments/procedures
- Study procedures
- o Serious adverse event reporting
- Study drug dosing
- Visit schedule/interval
- o Other

Every category will be kept in the summary even if it has 0 subjects. Subjects with more than 1 major protocol deviation will be counted only once in the total number of subjects with major protocol deviations. The following listing of all protocol deviations will be provided with deviation category, description, and a flag for major protocol deviation:

• All Protocol Deviations

#### 9. EFFICACY

All efficacy analyses will be performed using the Efficacy Evaluable Analysis Set, unless otherwise specified.

# 9.1. Primary Efficacy Endpoint and Analysis

#### 9.1.1. Primary Efficacy Endpoint

The primary efficacy endpoint is the incidence of CAR-T-associated neurotoxicity of any grade defined by CTCAE v5.0 by CAR-T Day +30. See Section 7.2.3.2 for the identification of the AE evaluations at the primary efficacy evaluation visit scheduled on CAR-T Day +30 to be used in the analysis. The actual number of efficacy evaluable subjects and the number of efficacy evaluable subjects who did not experience CAR-T-associated neurotoxicity of any grade by CAR-T Day +30 will be provided. The rate of no CAR-T-associated neurotoxicity of any grade will be estimated using the method of Koyama and Chen (2008), which incorporates the 2-stage design. The corresponding confidence interval (CI) and p-value will also be calculated using the method of Koyama and Chen (2008). If the actual Stage 2 sample size is the planned sample size, the null hypothesis will be rejected if 15 or more subjects with no CAR-T-associated neurotoxicity of any grade post-CAR-T-cell therapy by CAR-T Day +30 are observed in these 29 subjects. If the actual Stage 2 sample size is not the planned sample size, the method that takes both the planned and actual sample sizes into account for the 2-stage design will be used to calculate the rate of no CAR-T-associated neurotoxicity, the corresponding CI, and p-value (Koyama and Chen 2008); rejection of the null hypothesis after Stage 2 will be based on the p-value. The following summary will be provided:

• Analysis of the Incidence of CAR-T-associated Neurotoxicity of Any Grade Defined by CTCAE v5.0 by CAR-T Day +30 for All Efficacy Evaluable Subjects

The following listing of all CAR-T-associated neurotoxicity of any grade defined by CTCAE v5.0 by CAR-T Day +30 will be provided for all subjects enrolled at RP2D and having Yescarta infusion, with the start date of Yescarta administration/Study Day, the start date of the CAR-T-associated neurotoxicity/Study Day/CAR-T Day, the MedDRA High Level Group Term (HLGT) of the neurotoxicity, the grade of the neurotoxicity, a flag for being in the Efficacy Evaluable Analysis Set, and a flag for being in the Enrolled (RP2D) Analysis Set:

• All CAR-T-associated Neurotoxicity of Any Grade Defined by CTCAE v5.0 by CAR-T Day +30

For each subject who experienced CAR-T-associated neurotoxicity of any grade by CAR-T Day +30, all reported CAR-T-associated neurotoxicity events by CAR-T Day +30 will be included in this listing.

# 9.1.2. CTCAE v5.0 Grading of Neurotoxicity

The MedDRA HLGTs that are indicative of neurotoxicity are shown in Appendix 1. Each of these HLGTs is in the MedDRA SOC of either Nervous System Disorders or Psychiatric Disorders. The CTCAE v5.0 grading for AEs in the Nervous System Disorder and Psychiatric Disorder SOCs is shown in Appendix 2, and this will be used to grade events of neurotoxicity.

## 9.1.3. Analysis of the Primary Efficacy Endpoint

A Simon's design is usually indexed by 4 numbers that represent Stage 1 sample size  $(n_1)$ , Stage 1 critical value  $(R_1)$ , final sample size  $(n_t)$ , and final critical value  $(R_t)$ . Let  $X_1$  be the number of successes in Stage 1,  $X_2$  be the number of successes in Stage 2, and  $X_t$  be the total number of successes (ie,  $X_t = X_1 + X_2$ ), so  $X_1$  follows a binomial distribution with parameters  $n_1$  and  $n_2$  and  $n_3$  follows a binomial distribution with parameters  $n_2$  and  $n_3$  where  $n_2 = n_1 - n_2$  is the Stage 2 sample size. The rules for using the critical values,  $n_2$  and  $n_3$  are:

- If  $X_1 < R_1$ , the trial will be stopped for futility; otherwise, an additional sample will be taken until a total number of  $n_t$  subjects are obtained.
- Out of the  $n_t$  subjects, if  $X_t \ge R_t$ , efficacy is concluded by rejecting H<sub>0</sub>; otherwise, futility is concluded.

Therefore, for this study,  $n_1 = 10$ ,  $R_1 = 5$ ,  $n_t = 29$ , and  $R_t = 15$  (see Section 5.3).

If  $X_1 < R_1$  and futility is concluded in Stage 1, the p-value can be calculated as

$$P(X_1 \ge x_1 | p = p_0),$$

where  $x_1$  is the observed number of successes in Stage 1, and  $p_0$  is the probability of success under H<sub>0</sub>. For this study, the probability of success is the rate of no CAR-T-associated neurotoxicity and  $p_0 = 36\%$  (see Section 7.3). If the study continues to Stage 2, the p-value can be calculated as

$$\sum_{x_1=R_1}^{n_1} P(X_1=x_1|p=p_0)cp(x_1,x_2,n_2,p_0), \tag{1}$$

where  $cp(x_1, x_2, n_2, p_0) = P(X_2 \ge x_2 | X_1 = x_1, p = p_0)$ ,  $x_2$  is the observed number of successes in Stage 2 (ie,  $x_2 = x_t - x_1$ ), and  $x_t$  is the observed total number of successes. The term  $cp(x_1, x_2, n_2, p_0)$  can be called as the conditional p-value, which is the p-value of Stage 2 given the result of Stage 1. Under the situation that the actual Stage 2 is not the planned sample size,  $cp(x_1, x_2, n_2, p_0)$  in (1) will be replaced by  $A(x_1, n_2, p^*)$ , in order to be extended to the potential values of  $X_1$ ; therefore, the p-value can be calculated as

$$\sum_{x_1=R_1}^{n_1} P(X_1=x_1|p=p_0)A(x_1,n_2,p^*), \tag{2}$$

where  $A(x_1, n_2, p)$ , called the conditional power of Stage 2 given the results of Stage 1, can be calculated as

$$A(x_1, n_2, p) = \sum_{x_2 = R_2(x_1)}^{n_2} {n_2 \choose x_2} p^{x_2} (1 - p)^{(n_2 - x_2)},$$
 (3)

 $p^*$  is the solution of  $A(x_1, n_2, p^*) = cp(x_1, x_2, n_2, p_0)$ , and  $R_2(x_1) = R_t - x_1$  for  $R_1 \le x_1 < R_t$ , and 0 for  $R_t \le x_1$ .

To maintain consistency between hypothesis testing and CI, since Simon's design is used in the setting of 1-sided hypothesis testing, a 1-sided CI of the form  $(p_L, 1]$  will be calculated. With a type I error rate of 0.05, a 2-sided 90% CI will be calculated to obtain the lower bound for the 1-sided CI  $(p_L)$ . Using formula (1), a p-value can be calculated to test  $H_0$ :  $p \le p'_0$  for any  $p'_0$ . A 2-sided 90% CI is a collection of  $p'_0$  such that the corresponding p-value is within the interval of [0.05, 0.95]. If the Stage 2 sample size is not the planned sample size, formula (2) will be used instead to calculate of the CI.

The maximum likelihood estimator of p, denoted by  $\hat{p}$ , can be calculated as  $\hat{p} = x_t/n_t$ , if  $x_1 \ge R_1$  or  $\hat{p} = x_1/n_1$ , if  $x_1 < R_1$ , and has been shown to underestimate the true success probability in Simon's designs (Koyama and Chen 2008). Formula (1) with  $p = p'_0$  can be used to calculate the p-value to test  $H_0$ :  $p \le p'_0$  for any  $p'_0$ , as mentioned above. The value of  $p'_0$  that makes the p-value = 0.5 can be used as a reasonable estimate of p. If the Stage 2 sample size is not the planned sample size, formula (2) will be used instead to calculate of the point estimate of p.

The R functions that compute the p-value, point estimate and CI using the methods described above can be found using the following link:

http://biostat.mc.vanderbilt.edu/wiki/pub/Main/TatsukiRcode/twostage2018Web.R.

#### 9.1.4. Sensitivity Analyses

# 9.1.4.1. Sensitivity Analysis: Analysis of CAR-T-associated Neurotoxicity of Any Grade Defined by CTCAE v5.0 by CAR-T Day +30 for All Enrolled Subjects Treated at RP2D and Having Yescarta Infusion

The primary efficacy endpoint will be analyzed based on the Enrolled (RP2D) Analysis Set for this sensitivity analysis. The maximum likelihood estimate (MLE) for the rate of no CAR-T-associated neurotoxicity of any grade defined by CTCAE v5.0 by CAR-T Day +30 (ie, the sample proportion for subjects with no CAR-T-associated neurotoxicity of any grade defined by CTCAE v5.0 by CAR-T Day +30) will be calculated. The following summary will be provided:

 Analysis of the Incidence of CAR-T-associated Neurotoxicity of Any Grade Defined by CTCAE v5.0 by CAR-T Day +30 for All Enrolled Subjects Treated at RP2D and Having Yescarta Infusion

For the listing of all CAR-T-associated neurotoxicity of any grade corresponding to this sensitivity analysis, refer to the listing of All CAR-T-associated Neurotoxicity of Any Grade Defined by CTCAE v5.0 by CAR-T Day +30 specified in Section 9.1.1.

# 9.1.4.2. Sensitivity Analysis: Analysis of CAR-T-associated Neurotoxicity of Any Grade Defined by CTCAE v5.0 by CAR-T Day +30 for All Subjects Enrolled at RP2D and Having Yescarta Infusion

For this sensitivity analysis, subjects enrolled at RP2D who had Yescarta infusion but did not receive any defibrotide will be included, in addition to the subjects in the Enrolled (RP2D) Analysis Set. This analysis will be conducted using the same methods as the sensitivity analysis described in Section 9.1.4.1. The following summary will be provided:

 Analysis of the Incidence of CAR-T-associated Neurotoxicity of Any Grade Defined by CTCAE v5.0 by CAR-T Day +30 for All Subjects Enrolled at RP2D and Having Yescarta Infusion

For the listing of all CAR-T-associated neurotoxicity of any grade corresponding to this sensitivity analysis, refer to the listing of All CAR-T-associated Neurotoxicity of Any Grade Defined by CTCAE v5.0 by CAR-T Day +30 specified in Section 9.1.1.

If all subjects enrolled at RP2D are treated with at least 1 dose of defibrotide, this sensitivity analysis is the same as the sensitivity analysis specified in Section 9.1.4.1, and therefore will not be performed.

## 9.1.5. Subgroup Analyses

Not applicable.

# 9.2. Secondary Endpoints and Analyses

# 9.2.1. Secondary Efficacy Endpoint

# 9.2.1.1. Incidence of CAR-T-associated Neurotoxicity of Grade 3 or Greater Defined by CTCAE v5.0 by CAR-T Day +30

The MLE for the rate of no CAR-T-associated neurotoxicity of Grade 3 or greater defined by CTCAE v5.0 by CAR-T Day +30 (ie, the sample proportion for subjects with no CAR-T-associated neurotoxicity of Grade 3 or greater defined by CTCAE v5.0 by CAR-T Day +30) will be calculated. The following summary will be provided:

• Analysis of the Incidence of CAR-T-associated Neurotoxicity of Grade 3 or Greater Defined by CTCAE v5.0 by CAR-T Day +30 for All Efficacy Evaluable Subjects

For the listing of all CAR-T-associated neurotoxicity of Grade 3 or greater corresponding to this analysis, refer to the listing of All CAR-T-associated Neurotoxicity of Any Grade Defined by CTCAE v5.0 by CAR-T Day +30 specified in Section 9.1.1.

# 9.2.1.2. Incidence of CAR-T-associated Neurotoxicity (Any Grade and Grade 3 or Greater) according to the ASBMT Consensus Grading System by CAR-T Day +30

The MLE for the rate of no CAR-T-associated neurotoxicity of any grade (Grades 1, 2, 3 or 4) according to the ASBMT consensus grading system by CAR-T Day +30 (ie, the sample proportion for subjects with no CAR-T-associated neurotoxicity of any grade according to the ASBMT consensus grading system by CAR-T Day +30) will be calculated. The MLE for the rate of no CAR-T-associated neurotoxicity of Grade 3 or greater according to the ASBMT consensus grading system by CAR-T Day +30 (ie, the sample proportion for subjects with no CAR-T-associated neurotoxicity of Grade 3 or greater according to the ASBMT consensus grading system by CAR-T Day +30) will be calculated. See Section 7.2.3.1 for identification of the neurotoxicity evaluations at the primary efficacy evaluation visit scheduled on CAR-T Day +30 to be used in the analyses. There will be no hypothesis testing for the analysis of either of these secondary endpoints. The ASBMT consensus grading of CAR-T-associated neurotoxicity is provided in Appendix 3. The following summary will be provided:

 Analysis of the Incidence of CAR-T-associated Neurotoxicity according to the ASBMT Consensus Grading System by CAR-T Day +30 for All Efficacy Evaluable Subjects

including the following two sections:

- o Analysis of the incidence of CAR-T-associated neurotoxicity of any grade
- o Analysis of the incidence of CAR-T-associated neurotoxicity of Grade 3 or greater

The following listing of all CAR-T-associated neurotoxicity of any grade according to the ASBMT consensus grading system by CAR-T Day +30 will be provided for all efficacy evaluable subjects, with the start date of Yescarta administration/Study Day, the start date of the CAR-T-associated neurotoxicity/Study Day/CAR-T Day, the grades of ICE score, depressed level of consciousness, seizure, motor finding, and raised intracranial pressure/cerebral edema, and the grade of the neurotoxicity:

 All CAR-T-associated Neurotoxicity of Any Grade according to the ASBMT Consensus Grading System by CAR-T Day +30

For each subject who experienced CAR-T-associated neurotoxicity of any grade by CAR-T Day +30, all reported CAR-T-associated neurotoxicity events by CAR-T Day +30 will be included in this listing.

# 9.2.1.3. Incidence of CRS (Any Grade according to the ASBMT Consensus Grading System) by CAR-T Day +30

The MLE for the rate of no CRS of any grade (Grades 1, 2, 3 or 4) according to the ASBMT consensus grading system by CAR-T Day +30 (ie, the sample proportion for subjects with no CRS of any grade according to the ASBMT consensus grading system by CAR-T Day +30) will be calculated. See Section 7.2.3.1 for the identification of the CRS grading at the primary efficacy evaluation visit scheduled on CAR-T Day +30 to be used in the analysis. The grading of CRS by ASBMT criteria is provided in Appendix 4. The following summary will be provided:

• Analysis of the Incidence of CRS of Any Grade according to the ASBMT Consensus Grading System by CAR-T Day +30 for All Efficacy Evaluable Subjects

The following listing of all CRS of any grade according to the ASBMT consensus grading system by CAR-T Day +30 will be provided for all subjects enrolled at RP2D and having Yescarta infusion, with the start date of Yescarta administration/Study Day, the date of CRS assessment/Study Day/CAR-T Day, the grades of hypotension and hypoxia, a flag for being in the Efficacy Evaluable Analysis Set, and a flag for being in the Enrolled (RP2D) Analysis Set:

 All CRS of Any Grade according to the ASBMT Consensus Grading System by CAR-T Day +30

For each subject who experienced CRS of any grade by CAR-T Day +30, all reported CRS events by CAR-T Day +30 will be included in this listing.

# 9.2.1.4. Use of High Dose Steroid by CAR-T Day +30

The information regarding use of high dose steroid will be flagged on the Prior and Concomitant Medications page of the CRF. For the analyses of this secondary efficacy endpoint, use of high

dose steroid to treat CAR-T-associated neurotoxicity is the event of interest. The number of subjects who used high dose steroids by CAR-T Day +30 to treat CAR-T-associated neurotoxicity will be reported. The MLE for the proportion of subjects who use high dose steroids by CAR-T Day +30 to treat CAR-T-associated neurotoxicity (ie, the sample proportion for subjects who used high dose steroids by CAR-T Day +30 to treat CAR-T-associated neurotoxicity) will be calculated. For the subjects who used high dose steroids by CAR-T Day +30 to treat CAR-T-associated neurotoxicity, the time in days from the start of Yescarta administration to the start of high dose steroids, and the duration of use will be summarized separately using descriptive statistics. If use of high dose steroids is ongoing at the time of study completion, study withdrawal, or death, the date of study completion, study withdrawal, or death will be used to calculate the duration of use for the summary. The following summary will be provided:

 Analysis of Use Of High Dose Steroid by CAR-T Day +30 to Treat CAR-T-associated Neurotoxicity for All Efficacy Evaluable Subjects

The following listing of all incidence of high dose steroid use to treat CAR-T-associated neurotoxicity by CAR-T Day +30 will be provided for all efficacy evaluable subjects with the start date of Yescarta administration/Study Day, the start date/Study Day/CAR-T Day, ongoing (Yes or No), the end date, if not ongoing, dose (unit), frequency, and route:

• Use of High Dose Steroid by CAR-T Day +30 to Treat CAR-T-associated Neurotoxicity

All incidence of high dose steroid use to treat CAR-T-associated neurotoxicity by CAR-T Day +30 will be included in this listing.

# 9.2.2. Sensitivity Analyses

A sensitivity analysis will be performed for the following secondary efficacy endpoint: the incidence of CRS (any grade according to the ASBMT consensus grading system) by CAR-T Day +30 using the Enrolled (RP2D) Analysis Set. The analysis will be conducted using the same methods as described in Section 9.2.1.3. The following summary will be provided:

• Analysis of the Incidence of CRS of Any Grade according to the ASBMT Consensus Grading System by CAR-T Day +30 for All Enrolled Subjects at RP2D

For the listing of all CRS of any grade corresponding to this sensitivity analysis, refer to the listing of All CRS of Any Grade according to the ASBMT Consensus Grading System by CAR-T Day +30 specified in Section 9.2.1.3.

#### 9.2.3. Subgroup Analyses

Not applicable.

# 9.3. Exploratory Endpoints

## 9.3.1. Duration of Hospital Stay and ICU Stay

For the analyses of these endpoints, the following rules will be used to determine the hospitalization admission and discharge dates, and ICU admission and discharge dates under certain situations specified below:

- If the hospitalization admission date or ICU admission date is prior to the date of informed consent, use the date of informed consent as the hospitalization admission date or ICU admission date.
- If a subject is hospitalized or in the ICU at the time of study completion, study withdrawal, or death, use the date of study completion, study withdrawal, or death as the hospitalization discharge date or ICU discharge date.

The number of days for hospital stay will be calculated using the formula below:

**Days of hospital stay** = [Hospitalization discharge date] – [Hospitalization admission date] + 1.

If a subject is admitted to the hospital multiple times while on study, the number of days for hospital stay for this subject will be the sum of days of all hospital stays. The number of days for hospital stay will be summarized and presented using descriptive statistics. The number of days in ICU will be calculated using the formula below:

The number of days in ICU = [ICU discharge date] - [ICU admission date] + 1.

If a subject is admitted to ICU multiple times while on study, the number of days in ICU for this subject will be the sum of days of all ICU stays. The number of days in ICU will be summarized and presented using descriptive statistics. The following summary will be provided:

- Analysis of Duration of Hospital Stay and ICU Stay for All Efficacy Evaluable Subjects and the following sections will be included in the summary:
  - Hospital stay
  - o ICU stay

The following listing of all hospital stays will be provided with hospitalization admission date, hospitalization discharge date, was the subject admitted to the ICU (Yes or No), ICU admission date, and ICU discharge date:

• Duration of Hospital Stay and ICU Stay

For each subject, if there are multiple hospital stays, each hospital stage will be listed separately. For each hospital stay, if there is no ICU stay, ICU admission date and ICU discharge date will be left blank in the listing. If there is an ICU stay with no hospital stay, hospitalization admission date and hospitalization discharge date will be left blank in the listing. For one hospital stay, if there are multiple ICU stays, the information will be listed in the following format:

| Subject<br>Identifier/<br>Age/<br>Race | Hospitalization<br>Admission Date | Hospitalization<br>Discharge Date | Was the subject<br>admitted to the<br>ICU? | ICU Admission<br>Date | ICU Discharge<br>Date |
|---|---|---|---|---|---|
| 10011001/<br>17/<br>White | Hospitalization<br>Admission Date | Hospitalization<br>Discharge Date | Yes | ICU Admission<br>Date 1 | ICU Discharge<br>Date 1 |
| ,,,,,,,, | | | | ICU Admission<br>Date 2 | ICU Discharge<br>Date 2 |

# 9.3.2. Duration of CAR-T-associated Neurotoxicity by CTCAE v5.0

The following summaries will be provided:

- Analysis of Duration of CAR-T-associated Neurotoxicity of Any Grade Defined by CTCAE v5.0 for All Efficacy Evaluable Subjects
- Analysis of Duration of CAR-T-associated Neurotoxicity of Grade or Greater Defined by CTCAE v5.0 for All Efficacy Evaluable Subjects

For each of these analyses, the duration of CAR-T-associated neurotoxicity for each subject will be calculated in the following 2 ways:

- Method 1: duration is defined as the number of days between the start date of the first observed event and the end date of the last observed event.
- Method 2: duration is defined as the number of days between the start date of the first observed event and the end date of the last observed event, excluding the number of days in between on which no event was observed.

For the CAR-T-associated neurotoxicity that is ongoing at study completion, study withdrawal, or death, the date of study completion, study withdrawal or death will be used as the end date of that event.

#### 10. SAFETY

Safety analyses will be performed by dose level for Part 1 and for the phase 2 part of the study, using the Safety Analysis Set, unless otherwise specified. Note that since subjects treated at the RP2D in Part 1 will also be included in the phase 2 part under the 2-stage design, those subjects will be included in the summaries for both Part 1 and the phase 2 part of the study.

# 10.1. Exposure

#### 10.1.1. Extent of Exposure

A summary of defibrotide exposure will be provided using descriptive statistics:

Defibrotide Exposure by Study Phase

The following information will be included in the summary:

- Days of defibrotide exposure: number of days on which a subject received at least
   1 dose of defibrotide
- Total number of doses received
- o Total number of doses received before date of Yescarta
- o Total number of doses received on and after date of Yescarta
- o Number of doses per day before date of Yescarta:

[Total number of doses received before date of Yescarta] ÷ [Days of defibrotide exposure before date of Yescarta]

o Number of doses per day on and after date of Yescarta:

[Total number of doses received on and after date of Yescarta] ÷ [Days of defibrotide exposure on and after date of Yescarta]

Number of doses per day:

[Total number of doses received] ÷ [Days of defibrotide exposure]

- O Total exposure in mg: total amount of defibrotide received by a subject
- Daily dose in mg/day:

[Total exposure in mg] ÷ [Days of defibrotide exposure]

o Daily dose in mg/kg/day:

[Daily dose in mg/day] ÷ [Weight at baseline in kg]

The following listing of defibrotide administration will be provided, including the information regarding dose number per 24 hours, was dose given (Yes or No), start date/time, end date/time, dose per administration (unit), was defibrotide given as protocol specified time frame (Yes or No), and reason for delay:

• Defibrotide Administration
For the administration of defibrotide given with lymphodepletion chemotherapy, dose number per 24 hours is not applicable and will be specified as such in this listing.

#### **10.1.2.** Treatment Compliance

Not applicable.

#### 10.2. Adverse Events

Adverse events recorded in the CRF will be coded to SOC and PT using MedDRA 21.1. Investigators will assess the relatedness of each AE to defibrotide and to study procedures. The severity of AEs will be recorded using CTCAE, version 5.0.

Adverse events are graded by the investigator as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal). The severity grade of events for which the severity was not recorded will be categorized as "missing" for summaries and listings, and will be considered the least severe for the purposes of sorting for data presentation.

Treatment-related AEs for defibrotide are those for which investigators answer "Yes" to the question "Is this event related to study drug (Defibrotide)?" in the CRF. Events for which investigators do not record relationship to defibrotide will be considered as related to defibrotide for summary purpose (see Section 7.2.4.4). Listings will show treatment-relationship as missing. AEs for which "Yes" is marked for the question "Is this event related to study procedure?" in the CRF will be identified and included in AE listings.

Serious AEs are those for which investigators answers "Yes" to the question "Serious?" in the CRF. The clinical database will be reconciled with the SAE database before the final database lock.

A TEAE is defined as any event with a start date on or after the first dose date and up to 30 days after the last dose of defibrotide, or any ongoing event that worsens in severity after the first dose date and up to 30 days after the last dose of defibrotide. Only TEAEs with the onset date through the end of the AE reporting period (30 days after the last dose of defibrotide) will be included in the summaries unless otherwise specified. For the purpose of determining treatment-emergent, incomplete and missing AE start dates will be imputed as specified in Section 7.2.4.1.

See Section 7.2.3.2 for the identification of the AE evaluations at the final safety follow-up visit scheduled on CAR-T Day +37 to be included in the analyses.

#### **10.2.1.** Dose-limiting Toxicities

During Part 1 of the study, all TEAEs that occur from the start of the first dose of defibrotide up to 7 days after the last dose of defibrotide will be screened for DLT. The final determination of DLTs will then be made by the SAC from TEAEs considered to have a causal relationship to defibrotide. As an exception, all bleeding TEAEs, regardless of relationship to defibrotide will be evaluated by the SAC as potential DLTs. Because all hemorrhagic events are considered adverse drug reactions of defibrotide, the SAC will review any grade (per CTCAE v5.0) of intracranial hemorrhage and any other hemorrhage of Grade 2 or greater. The SAC will also review all nonhemorrhagic TEAEs of Grade 3 or greater as possible DLTs. Of note, CAR-T-associated neurotoxicity is not a DLT. The number of subjects with DLTs for each cohort in Part 1 will be summarized by cohort using the Safety Analysis Set. The following summary will be provided:

• DLTs by Cohort for Part 1

The following listing of all DLTs for Part 1 will be provided with subject identifier, dose level, SOC, PT, start date, end date, severity grade, seriousness, relationship to defibrotide, relationship to a study procedure, action taken, and outcome of the AE:

• All DLTs for Part 1

#### 10.2.2. Adverse Events

The following summaries of AEs will be provided for all subjects in the Safety Analysis Set:

- TEAEs by PT and by Study Phase
- Serious TEAEs by SOC and PT and by Study Phase
- Treatment-related TEAEs by SOC and PT and by Study Phase
- Serious Treatment-related TEAEs by SOC and PT and by Study Phase
- TEAEs Leading to Defibrotide Discontinuation by SOC and PT and by Study Phase
- Treatment-related TEAEs Leading to Defibrotide Discontinuation by SOC and PT and by Study Phase
- TEAEs Leading to Death by SOC and PT and by Study Phase
- Treatment-related TEAEs Leading to Death by SOC and PT and by Study Phase
- TEAEs by SOC and PT, by Maximum Severity and by Study Phase
- Treatment-related TEAEs by SOC and PT, by Maximum Severity and by Study Phase

Treatment-emergent AEs will be summarized by PT, sorted in descending order of incidence for the phase 2 part of the study. The other AE summaries will be provided by SOC and PT, and SOCs will be ordered alphabetically, with PTs within an SOC sorted in descending order of incidence for the phase 2 part of the study. If a subject has more than 1 AE within a PT, the subject is counted only once at the maximum severity; if a subject has more than 1 AE within an SOC, the subject is counted once at the maximum severity when reporting results for that SOC.

Additionally, the following TEAE summaries for public disclosure will be provided:

- Summary of Treatment-emergent Serious Adverse Events (for Public Disclosure)
- Summary of Treatment-emergent Non-serious Adverse Events Occurring in Greater Than 5% of Subjects

The following listings will be provided with subject identifier, study part, SOC, PT, start date, end date, severity grade, seriousness, relationship to defibrotide, relationship to a study procedure, action taken, and outcome of the AE:

- All AEs
- AEs Leading to Death
- CTCAE Grade 3 to 5 AEs
- Serious AEs

#### **10.2.3.** Adverse Events of Special Interest

As TEAEs of special interest, bleeding events will be summarized by SOC and PT. The MedDRA 21.1 Standardised MedDRA Query (SMQ) Haemorrhage terms (excluding laboratory terms) will be used to search for bleeding events and is provided in Appendix 5. The following summary will be provided:

• TEAEs of Special Interest: Bleeding by SOC and PT and by Study Phase

System organ classes will be ordered alphabetically, with PTs within an SOC sorted in descending order of incidence in the defibrotide prophylaxis arm. If a subject has more than 1 TEAE of special interest within a PT, the subject is counted only once at the maximum severity; if a subject has more than 1 TEAE of special interest within an SOC, the subject is counted once at the maximum severity when reporting results for that SOC.

The following listing of all TEAEs of special interest: bleeding will be provided with subject identifier, study part, SOC, PT, start date, end date, severity grade, seriousness, relationship to defibrotide, relationship to a study procedure, action taken, and outcome of the AE:

TEAEs of Special Interest: Bleeding

#### 10.2.4. Summary of Adverse Events

The following summary of AEs will be provided:

• Summary of Adverse Events by Study Phase and Overall

The following information will be included in the summary: the numbers of subjects with at least 1 TEAE, the numbers of subjects with at least 1 serious TEAE, the numbers of subjects with at least 1 treatment-related TEAE, the numbers of subjects with at least 1 serious treatment-related TEAE, the numbers of subjects with at least 1 TEAE of Grade 3 or greater, the numbers of subjects with at least 1 treatment-related TEAE of Grade 3 or greater, the numbers of subjects with TEAEs leading to defibrotide discontinuation, the numbers of subjects with treatment-related TEAEs leading to death, the numbers of subjects with treatment-related TEAEs leading to death, and the numbers of subjects with at least 1 TEAE of special interest: bleeding.

### 10.3. Laboratory Assessments

For the following laboratory tests:

- chemistry: blood urea nitrogen, calcium, chloride, direct bilirubin, indirect bilirubin, magnesium, potassium, phosphorus, sodium, total bilirubin, and total protein
- hematology: hematocrit, mean corpuscular volume, basophils (absolute and relative), eosinophils (absolute and relative), relative lymphocyte count, monocytes (absolute and relative), relative neutrophil count, bands (absolute and relative), and blast (absolute and relative)
- coagulation: activated partial thromboplastin time, and international normalized ratio a shift table of post-baseline results (with respect to the normal range value) from baseline will be provided for each type of laboratory tests:

- Shift Table from Baseline of Selected Laboratory Results with Respect to the Normal Range by Study Phase: Chemistry
- Shift Table from Baseline of Selected Laboratory Results with Respect to the Normal Range by Study Phase: Hematology
- Shift Table from Baseline of Selected Laboratory Results with Respect to the Normal Range by Study Phase: Coagulation

For each laboratory test, the shift table will include change in normal range value from baseline for the worst post-baseline case. Lab values at unscheduled visits, if any, will also be considered, and subjects with both abnormal low and high post-baseline values will be counted twice.

For the following laboratory tests:

- chemistry: alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, calcium, creatinine, glucose, magnesium, potassium, sodium, and total bilirubin
- hematology: hemoglobin, platelet count, white blood cell count, absolute lymphocyte count, and absolute neutrophil count

a shift table of post-baseline results (in CTCAE v5.0 grade) from baseline will be provided for each type of laboratory tests:

- Shift Table in CTCAE v5.0 Grade from Baseline of Selected Laboratory Results by Study Phase: Chemistry
- Shift Table in CTCAE v5.0 Grade from Baseline of Selected Laboratory Results by Study Phase: Hematology

For each laboratory test, the shift table will include change in CTCAE v5.0 grade from baseline for the worst post-baseline case. Lab values at unscheduled visits, if any, will also be considered.

A listing of abnormal post-baseline lab values for each type of laboratory tests will be provided with specimen collection date/Study Day, test name, result (unit), corresponding normal ranges, and reference range flag:

- Abnormal Post-baseline Laboratory Values: Chemistry
- Abnormal Post-baseline Laboratory Values: Hematology
- Abnormal Post-baseline Laboratory Values: Urinalysis
- Abnormal Post-baseline Laboratory Values: Coagulation

### 10.4. Vital Signs

For systolic blood pressure, diastolic blood pressure, pulse rate, respiratory rate, and body temperature, a shift table of post-baseline results (with respect to the normal range value) from baseline will be provided:

• Shift Table from Baseline of Selected Vital Signs with Respect to the Normal Range by Study Phase

For each vital sign listed above, the shift table will include change in normal range value from baseline for the worst post-baseline case. Vital signs at unscheduled visits, if any, will also be considered, and subjects with both abnormal low and high post-baseline values will be counted twice.

A listing abnormal post-baseline vital sign values will be provided with date of measurement/Study Day, test name, body temperature measurement method (for body temperature only), and result (unit):

• Abnormal Post-baseline Vital Signs

In order to create the shift table and the listing, the following values are considered to represent abnormal vital signs:

- Systolic blood pressure < 60 or > 160 mmHg
- Diastolic blood pressure < 50 or > 100 mmHg
- Pulse rate < 40 or > 120 beats per minute
- Respiratory rate < 10 or > 40 breaths per minute
- Temperature < 36 or > 39 degrees Centigrade

#### 10.5. Lymphoma Response

Investigator assessed outcome of Yescarta response will be summarized with the following categories: complete response, partial response, stable disease, progressive disease, and not evaluable. For the purpose of the summary, if lymphoma response information is missing for a subject, the subject will be considered to have had progressive disease (Section 7.2.4.5). The following summary will be provided:

Lymphoma Response by Study Phase

The following listing of lymphoma response will be provided with subject identifier, study part, date of overall response/Study Day/CAR-T Day, overall response, was a PET/CT scan performed (Yes or No), date of PET/CT scan and result (if Yes to was a PET/CT scan performed), was a bone marrow evaluation performed (Yes or No), date of bone marrow evaluation, bone marrow type and was the bone marrow involved with lymphoma (if Yes to was a bone marrow evaluation performed):

• Lymphoma Response

#### 11. PHARMACOKINETIC ANALYSES

#### 11.1. General Considerations

Some minor modifications may be necessary to the planned design of tables, figures, and listings to accommodate data collected during the actual study conduct.

Quantitative variables will be summarized using descriptive statistics (sample size, arithmetic mean, standard deviation, coefficient of variation, median, minimum, and maximum). Geometric statistics (mean and standard deviation) will be included for PK concentrations and parameters, where applicable.

All defibrotide concentration data will be reported and analyzed with the same precision as the source data provided by the bio-analytical laboratory regardless of how many significant figures or decimals the data carry. Derived PK parameters will be rounded for reporting purposes in listings. The rounded derived PK parameters will be considered the source data for the calculation of descriptive statistics and other statistical analysis. For most derived PK parameters, 3 significant digits will be used as the standard rounding procedure, with the following exceptions:

- Parameters directly derived from source data (eg, maximum defibrotide concentration [C<sub>max</sub>]) will be reported and analyzed with the same precision as the source data.
- Parameters derived from actual elapsed sample collection times (eg, time to maximum activity [T<sub>max</sub>]) will be reported with the same precision as the actual elapsed sampling time value of the source data.

For the reporting of descriptive statistics, the arithmetic and geometric means and standard deviations will be presented with precision of 1 digit more than the source data. The minimum, median, and maximum will be presented with the same precision as the source data. Coefficients of variation will always be reported with 1 decimal place.

#### 11.2. Defibrotide Plasma Concentrations

Analyses specified in this section will be performed using the PK Analysis Set.

For each dose level, the defibrotide plasma concentrations will be reported by Nominal Time Point (prior to defibrotide infusion, and 1, 2, 4, 6 and 24 hours post start of defibrotide infusion on CAR-T Day -5; prior to defibrotide infusion, and 2 and 4 hours post start of defibrotide infusion on CAR-T Day 0 and CAR-T Day +7), using descriptive statistics as described in Section 11.1. Concentrations that are below the limit of quantitation (BLQ) will be treated as a numeric value of 0, and the associated geometric statistics will be designated and reported as not done. The following summary will be provided:

• Defibrotide Plasma Concentrations by Dose Level and Nominal Time Point on CAR-T Day -5, CAR-T Day 0 and CAR-T Day +7

Figures of individual and arithmetic mean defibrotide concentration-time profiles ( $\pm$  standard deviation, as appropriate) using Nominal Time Points (prior to defibrotide infusion, and 1, 2, 4, 6 and 24 hours post start of defibrotide infusion on CAR-T Day -5) will be presented on linear and semi-logarithmic scales by dose level for the CAR-T Day -5 visit. For graphing purposes, the BLQ

values will be considered as missing and, if applicable, 2 neighboring values will be connected. The following figures will be provided:

- Mean Defibrotide Plasma Concentration-time Profile on Linear Scale following Defibrotide Infusion on CAR-T Day -5
- Mean Defibrotide Plasma Concentration-time Profile on Semi-logarithmic Scale following Defibrotide Infusion on CAR-T Day -5

A listing of all defibrotide plasma concentrations will be provided:

• Defibrotide Plasma Concentrations

#### 11.3. Defibrotide Pharmacokinetic Parameters

Analyses specified in this section will be performed using the PK Evaluable Analysis Set.

Subjects with partial defibrotide concentrations data, protocol violations or events with the potential to affect PK will be evaluated on a case-by-case basis to determine if sufficient data are available for reliable estimation of PK parameters. PK parameters will be calculated for the CART Day -5 visit as data permit.

The defibrotide plasma PK parameters will be calculated using the standard non-compartmental analysis methods according to current working practices and Phoenix WinNonlin (Certara USA, Inc., v6.3 or higher).

All calculations of non-compartmental parameters will be based on actual sampling times for the analysis, but all pre-dose times will be assigned a numerical value of 0 to prevent overestimation of the AUC.

Defibrotide plasma concentrations that are BLQ or missing will be handled the following way:

- Pre-dose sample concentrations that are BLQ or missing will be assigned a numerical value of 0.
- Any other BLQ value will be assigned a value of 0 if they precede quantifiable samples in the initial portion of the profile.
- A BLQ value that occurs between quantifiable data points, especially prior to C<sub>max</sub>, will be evaluated to determine if an assigned value of 0 makes sense, or if exclusion of the data (flagged in the data and identified to be treated as missing) is warranted.
- Following C<sub>max</sub>, the BLQ values embedded between 2 quantifiable data points will be treated as missing when calculating PK parameters.
- If a BLQ value occurs at the end of the collection interval (after the last quantifiable activity), it will be set to 0.
- If consecutive BLQ values are followed by quantifiable values in the terminal portion
  of the concentration curve, these quantifiable values will be excluded from the PK
  analysis by setting them to missing, unless otherwise warranted by the
  concentration-time profile.

Where possible, the following PK parameters will be determined from defibrotide plasma concentrations for the CAR-T Day -5 visit:

| C <sub>max</sub> | Maximum defibrotide plasma concentration, obtained directly from the observed data |
|---|---|
| T <sub>max</sub> | Time of maximum defibrotide concentration (in hours), obtained directly from the observed data |
| C <sub>last</sub> | The last quantifiable defibrotide concentration, obtained directly from observed data |
| T <sub>last</sub> | Time of the last quantifiable defibrotide concentration (in hours), obtained directly from the observed data |
| AUC <sub>0-t</sub> | Area under the defibrotide concentration-time curve in the sampled matrix from 0 (pre-dose) to time of last quantifiable defibrotide concentration at time "t" |
| AUC <sub>0-inf</sub> | Area under the defibrotide plasma concentration-time curve from 0 (pre-dose), extrapolated to infinity by addition of the last quantifiable concentration divided by the elimination rate constant to $AUC_{0-t}$ : $AUC_{0-t} + C_{last} / \lambda_z$ |
| $\lambda_z \left( k_{el} \right)$ | Apparent terminal elimination rate constant (in 1/hour), determined by linear regression of the terminal points of the log-linear defibrotide concentration-time curve |
| | Visual assessment will be used to identify the terminal linear phase of the defibrotide concentration-time profile. A minimum of 3 data points will be used for the determination. |
| t <sub>1/2</sub> | Terminal elimination half-life (in hours): $ln(2) / \lambda_z$ |
| CL | Systemic clearance after intravenous dosing, calculated as dose divided by AUC <sub>0-inf</sub> |
| V <sub>ss</sub> | Estimate of the volume of distribution at steady state following intravenous dosing: $MRT_{0-inf} \times CL$ , where $MRT_{0-inf}$ is mean residence time extrapolated to infinity |

All AUC parameters will be calculated using Linear trapezoidal / Linear Interpolation trapezoidal summation. The minimum requirement for the calculation of AUC will be the inclusion of at least 3 consecutive plasma concentrations above the lower limit of quantification, with at least 1 of these concentrations following  $C_{\text{max}}$ .

The following PK parameters will be calculated for diagnostic or parameter derivation purposes and listed, but will not be summarized.

| $t_{1/2}$ , Interval | The time interval (in hours) of the log-linear regression to determine $\lambda_z$ . |
|---|---|
| | The $t_{1/2}$ will be estimated over a time period of at least 2 half-lives, where |
| | possible. Where a $t_{1/2}$ is estimated over a time period of less than 2 half-lives, it |

| | may be flagged in the data listings at the discretion of the Pharmacokineticist, and the robustness of the value will be discussed in the CSR. |
|---|---|
| t <sub>1/2</sub> , N | Number of data points included in the log-linear regression analysis to determine $\lambda_z$ |
| | A minimum of 3 data points will be used for determination. |
| Rsq,<br>adjusted | Goodness of fit statistic for calculation of $\lambda_z$ |
| | A value of $\geq 0.8$ for the adjusted R-squared value will be used as the criterion for the reliable estimation of $\lambda_z$ and reporting of the $t_{1/2}$ . If the adjusted R-squared value does not meet this criterion for a given subject the $t_{1/2}$ , AUC <sub>0-inf</sub> , CL, and $V_{ss}$ will be listed but not included in the descriptive statistics. |
| %AUC <sub>extr</sub> | Percentage of AUC <sub>0-inf</sub> obtained by extrapolation: [(C <sub>last</sub> / $\lambda_z$ ) / AUC <sub>0-inf</sub> × 100] |
| | If %AUC <sub>extr</sub> is greater than 20% of AUC <sub>0-inf</sub> , then AUC <sub>0-inf</sub> , CL, and V <sub>ss</sub> will be listed but not included in summary statistics. |
| AUMClast | Area under the first moment curve (AUMC) from 0 (pre-dose) to time of last quantifiable defibrotide concentration at time "t" |
| AUMC <sub>0-inf</sub> | Area under the first moment curve extrapolated to infinity, based on the last observed concentration, calculated as $AUMC_{last} + \left(T_{last} \times C_{last}\right) / \lambda_z + C_{last} / \lambda_z$ |
| MRT <sub>0-inf</sub> | Mean residence time extrapolated to infinity, calculated for infusion models as $(AUMC_{0-inf} / AUC_{0-inf}) - TI / 2$ , where TI is infusion time |

All PK parameters will be summarized by dose level for the CAR-T Day -5 visit using descriptive statistics as described in Section 11.1. Geometric mean will not be calculated for  $T_{max}$  and  $T_{last}$ . The following summaries will be provided:

• Defibrotide Plasma Pharmacokinetic Parameters by Dose Level on CAR-T Day -5

A listing of all generated individual PK parameters will be provided:

• Defibrotide Plasma Pharmacokinetic Parameters on CAR-T Day -5

# 12. PHARMACODYNAMIC ANALYSES

Not applicable.

#### 13. **COVID-19**

Comments identifying missed visits, missed assessments, study drug discontinuation, and/or study participation termination due to COVID-19 will be captured in EDC. Additionally, comments will be captured in EDC if a visit is performed as a remote voice or video visit. Comments will specify if the study disruption was due to acquiring COVID-19 or due to other COVID-19 restrictions.

The following listing will be provided and will include all subjects affected by the COVID-19 related study disruption by unique subject number identifier and by investigational site, and a description of how the individual's participation was altered:

• Subjects Impacted by the COVID-19 Pandemic

#### REFERENCES

Lee DW, Santomasso BD, Locke FL, et al. ASBMT consensus grading for cytokine release syndrome and neurological toxicity associated with immune effector cells. Biol Blood Marrow Transplant 2019; 25(4): 625–638.

Cheson BD, Ansell S, Schwartz L, et al. Refinement of the Lugano Classification lymphoma response criteria in the era of immunomodulatory therapy. Blood 2016; 128(2): 2489-2496.

Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials 1989; 10(1): 1-10.

Neelapu SS, Locke FL, Bartlett NL, et al. Axicabtagene ciloleucel CAR T-cell therapy in refractory large B-cell lymphoma. N Engl J Med 2017; 377(26): 2531-2544.

Koyama T, Chen H. Proper inference from Simon's two-stage designs. Stat Med 2008; 27(16): 3145-3154.

Topp MS, Gökbuget N, Stein AS, et al. Safety and activity of blinatumomab for adult patients with relapses or refractory B-precursor acute lymphoblastic leukaemia: a multicentre, single-arm, phase 2 study. Lancet Oncol 2015; 16(1): 57-66.

# APPENDIX 1. MEDDRA HIGH LEVEL GROUP TERMS INDICATIVE OF NEUROTOXICITY

The high-level group terms that are indicative of neurotoxicity include (Topp et al. 2015):

Cranial nerve disorders

Deliria, including confusion

Disturbances in thinking and perception

Encephalopathies

Mental impairment disorders

Movement disorders, including Parkinsonism

Neurologic disorders not elsewhere classified (NEC)

Neuromuscular disorders

Personality disorders and disturbances in behavior

Psychiatric disorders NEC

Seizures, including subtypes

# APPENDIX 2. CTCAE VERSION 5.0 GRADING FOR NERVOUS SYSTEM DISORDERS AND PSYCHIATRIC DISORDERS

The severity of neurotoxicity events (defined in Appendix 1) should be based on CTCAE v5.0.

| Nervous system disord | lers | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| CTCAE Term | 1 | 2 | 3 | 4 | 5 |
| Abducens nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | d by dysfunction of the abducens n | erve (sixth cranial nerve). | | | |
| Accessory nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | d by dysfunction of the accessory n | erve (eleventh cranial nerve). | ' | | |
| Acoustic nerve disorder NOS | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | d by dysfunction of the acoustic ne | rve (eighth cranial nerve). | T | T | 1 |
| Akathisia | Mild restlessness or increased motor activity | Moderate restlessness or increased motor activity; limiting instrumental ADL | Severe restlessness or increased motor activity; limiting self care ADL | - | - |
| Definition: A disorder characterize | d by an uncomfortable feeling of in | ner restlessness and inability to stay | still; this is a side effect of some ps | ychotropic drugs. | |
| Amnesia | Mild; transient memory loss | Moderate; short term memory loss; limiting instrumental ADL | Severe; long term memory loss; limiting self care ADL | - | - |
| Definition: A disorder characterize | d by systematic and extensive loss of | of memory. | | | |
| Anosmia | Present | - | - | - | - |
| Definition: A disorder characterize | ed by a change in the sense of smell. | ' | ' | ' | ' |
| Aphonia | - | - | Voicelessness; unable to speak | - | - |
| Definition: A disorder characterize | d by the inability to speak. It may re | esult from injuries to the vocal cords | or may be functional (psychogenic | ). | |
| Arachnoiditis | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | d by inflammation of the arachnoid | membrane and adjacent subarachi | noid space. | | |
| Ataxia | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; mechanical assistance indicated | - | - |
| Definition: A disorder characterize | d by lack of coordination of muscle | movements resulting in the impairr | nent or inability to perform volunta | ry activities. | |
| Brachial plexopathy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | d by regional paresthesia of the bra | chial plexus, marked discomfort and | d muscle weakness, and limited mo | vement in the arm or hand. | |
| Central nervous system necrosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms;<br>corticosteroids indicated | Severe symptoms; medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | d by a necrotic process occurring in | the brain and/or spinal cord. | | | |
| Cerebrospinal fluid leakage | Post-craniotomy:<br>asymptomatic; Post-lumbar<br>puncture: transient headache;<br>postural care indicated | Post-craniotomy: moderate symptoms; medical intervention indicated; Post-lumbar puncture: persistent moderate symptoms; blood | Severe symptoms; medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ।<br>d by loss of cerebrospinal fluid into | patch indicated the surrounding tissues. | 1 | 1 | İ |

| Nervous system disor | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| CTCAE Term | 1 | 2 | 3 | 4 | 5 |
| Cognitive disturbance | Mild cognitive disability; not interfering with work/school/life performance; specialized educational services/devices not indicated | Moderate cognitive disability;<br>interfering with<br>work/school/life performance<br>but capable of independent<br>living; specialized resources on<br>part time basis indicated | Severe cognitive disability;<br>significant impairment of<br>work/school/life performance | - | - |
| Definition: A disorder characteriz | ed by a conspicuous change in cogni | | | | |
| Concentration impairment | Mild inattention or decreased level of concentration | Moderate impairment in attention or decreased level of concentration; limiting instrumental ADL | Severe impairment in attention<br>or decreased level of<br>concentration; limiting self care<br>ADL | - | - |
| | ed by a deterioration in the ability to | | | | |
| Depressed level of consciousness | Decreased level of alertness | Sedation; slow response to<br>stimuli; limiting instrumental<br>ADL | Difficult to arouse | Life-threatening consequences; coma; urgent ntervention indicated | Death |
| Definition: A disorder characteriz | ed by a decrease in ability to perceiv | e and respond. | | | |
| Dizziness | Mild unsteadiness or sensation of movement | Moderate unsteadiness or sensation of movement; limiting instrumental ADL | Severe unsteadiness or<br>sensation of movement;<br>limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a disturbing sensation of lighth | eadedness, unsteadiness, giddines | s, spinning or rocking. | T | |
| Dysarthria | Mild slurred speech | Moderate impairment of articulation or slurred speech | Severe impairment of articulation or slurred speech | - | - |
| Definition: A disorder characteriz | ed by slow and slurred speech result | ing from an inability to coordinate t | he muscles used in speech. | | |
| Dysesthesia Definition: A disorder characteriz | Mild sensory alteration ed by distortion of sensory perceptic | Moderate sensory alteration; limiting instrumental ADL | Severe sensory alteration;<br>limiting self care ADL | - | - |
| Dysgeusia | Altered taste but no change in | Altered taste with change in | _ | _ | _ |
| o y secusion | diet | diet (eg, oral supplements);<br>noxious or unpleasant taste;<br>loss of taste | | | |
| Definition: A disorder characteriz | ed by abnormal sensual experience v | with the taste of foodstuffs; it can b | e related to a decrease in the sense | of smell. | |
| Dysphasia<br>Definition: A disorder characteriz | Awareness of receptive or expressive characteristics; not impairing ability to communicate ed by impairment of verbal commun | Moderate receptive or expressive characteristics; impairing ability to communicate spontaneously ication skills, often resulting from b | Severe receptive or expressive characteristics; impairing ability to read, write or communicate intelligibly rain damage. | | - |
| Edema cerebral | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by swelling due to an excessive ac | ccumulation of fluid in the brain. | | | |
| Encephalopathy | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a pathologic process involving | the brain. | | | |
| Extrapyramidal disorder | Mild involuntary movements | Moderate involuntary<br>movements; limiting<br>instrumental ADL | Severe involuntary<br>movements or torticollis;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz<br>Facial muscle weakness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength of t | he facial muscles. | | | |
| Facial nerve disorder | Asymptomatic; clinical or diagnostic observations only; | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |

| | Crada | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| CTCAE Term | 1 | 2 | 3 | 4 | 5 |
| Glossopharyngeal nerve | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | Life-threatening | Death |
| disorder | diagnostic observations only; | instrumental ADL | care ADL | consequences; urgent | |
| | intervention not indicated | | | intervention indicated | |
| Definition: A disorder characteri | zed by dysfunction of the glossophary | /ngeal nerve (ninth cranial nerve). | | Т | ı |
| Guillain-Barre syndrome | Mild symptoms | Moderate symptoms; | Severe symptoms; limiting self | Life-threatening | Death |
| | | limiting instrumental | care ADL | consequences; urgen | |
| | | ADL | | intervention indicated; | |
| | | | | intubation | |
| Definition: A disorder characteri | zed by the body's immune system att | acking the peripheral nervous syste | em causing ascending paralysis. | | ı |
| Headache | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | | instrumental ADL | ADL | | |
| Definition: A disorder characteri | zed by a sensation of marked discomi | fort in various parts of the head, no | t confined to the area of distribution | of any nerve. | |
| Hydrocephalus | Asymptomatic; clinical or | Moderate symptoms; | Severe symptoms or | Life-threatening | Death |
| | diagnostic observations only; | intervention not indicated | neurological deficit; | consequences; urgent | |
| | intervention not indicated | | intervention indicated | intervention indicated | |
| Definition: A disorder characteri | zed by an abnormal increase of cereb | rospinal fluid in the ventricles of th | e brain. | T | |
| Hypersomnia | Mild increased need for sleep | Moderate increased need for | Severe increased need for | - | - |
| | | sleep | sleep | | |
| Definition: A disorder characteri | zed by excessive sleepiness during the | e daytime. | | | |
| Hypoglossal nerve disorder | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| | diagnostic observations only; | instrumental ADL | care ADL | | |
| | intervention not indicated | | l | | |
| Definition: A disorder characteri | zed by dysfunction of the hypoglossa | nerve (twelfth cranial nerve). | | T | |
| Intracranial hemorrhage | Asymptomatic; clinical or | Moderate symptoms; medical | Ventriculostomy, ICP | Life-threatening | Death |
| | diagnostic observations only; | intervention indicated | monitoring, intraventricular | consequences; urgent | |
| | intervention not indicated | | thrombolysis, or operative | intervention indicated | |
| | | | intervention indicated | | |
| Definition: A disorder characteri | zed by bleeding from the cranium. | T | | | |
| Ischemia cerebrovascular | Asymptomatic; clinical or | Moderate symptoms | - | - | - |
| | diagnostic observations only; | | | | |
| | intervention not indicated | | | | |
| Definition: A disorder characteri | zed by a decrease or absence of bloo | d supply to the brain caused by ob | struction (thrombosis or embolism) | of an artery resulting in neurological | al |
| damage. | | T | | | |
| Lethargy | Mild symptoms; reduced | Moderate symptoms; limiting | - | - | - |
| | alertness and awareness | instrumental ADL | | | |
| Definition: A disorder characteri | zed by a decrease in consciousness ch | naracterized by mental and physical | inertness. | T. | |
| Leukoencephalopathy | Asymptomatic; small focal | Moderate symptoms; focal | Severe symptoms; extensive | Life-threatening consequences; | Death |
| | T2/FLAIR hyperintensities; | T2/FLAIR hyperintensities, | T2/FLAIR hyperintensities, | extensive T2/FLAIR | |
| | involving periventricular white | involving periventricular white | involving periventricular white | hyperintensities, involving | |
| | matter or <1/3 of susceptible | matter extending into centrum | matter involving 2/3 or more of | periventricular white matter | |
| | areas of cerebrum +/- mild | semiovale or involving 1/3 to | susceptible areas of cerebrum | involving most of susceptible | |
| | increase in subarachnoid space | 2/3 of susceptible areas of | | areas of cerebrum | |
| | (SAS) and/or mild | cerebrum +/- moderate | +/- moderate to severe | | |
| | ventriculomegaly | increase in SAS and/or | increase in SAS and/or | +/- moderate to severe | |
| | | moderate ventriculomegaly | moderate to severe | increase in SAS and/or | |
| Definition: A disorder characteri | ed by diffuse reactive astrocytosis w | I<br>ith multiple areas of necrotic foci w | ventriculomegaly ithout inflammation. | moderate to severe | I |
| Memory impairment | Mild memory impairment | Moderate memory | Severe memory impairment; | _ | _ |
| y impanificht | a memory impairment | impairment; limiting | limiting self care ADL | | |
| | | instrumental ADL | | | |
| Definition: A disorder characteri | zed by a deterioration in memory fun | | • | ı | |
| Vieningismus | Mild symptoms | Moderate symptoms; limiting | Severe symptoms; limiting self | Life-threatening | Death |
| - '0' | | instrumental ADL | care ADL | consequences; urgent | |
| | | | | intervention indicated | |
| | zed by neck stiffness, headache, and | photophobia resulting from irritatio | on of the cerebral meninges. | • | • |
| Definition: A disorder characteri | | | | | |
| Definition: A disorder characteri Movements involuntary | Mild symptoms | Moderate symptoms; limiting | Severe symptoms; limiting self | _ | |

| Nervous system disord | iers | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| CTCAE Term | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characterize | ed by uncontrolled and purposeless | movements. | | | |
| Muscle weakness left-sided | Symptomatic; perceived by | Symptomatic; evidence | Limiting self care ADL | - | - |
| | patient but not evidence | on physical exam; | | | |
| | on physical exam | limiting instrumental | | | |
| Definition: A disorder characteriz | ed by a reduction in the strength of | the muscles on the left side of the | body. | | |
| Muscle weakness right-sided | Symptomatic; perceived by | Symptomatic; evidence | Limiting self care ADL | - | - |
| | patient but not evidence | on physical exam; | | | |
| | on physical exam | limiting instrumental | | | |
| Definition: A disorder characteriz | ed by a reduction in the strength of | the muscles on the right side of the | e body. | | |
| March and a sector | A | Mandamata, minimal | Carrage and and the significant | 116- About to the | D41 |
| Myasthenia gravis | Asymptomatic or mild | Moderate; minimal, | Severe or medically significant | Life-threatening | Death |
| | symptoms; clinical or diagnostic observations | local or noninvasive intervention indicated; | but not immediately life-threatening; | consequences; urgent intervention indicated | |
| | only; intervention not | limiting age-appropriate | hospitalization or prolongation | intervention indicated | |
| | indicated | instrumental ADL | of existing hospitalization | | |
| | marcacca | Janamental ADE | indicated; limiting self care ADL | | |
| Definition: A disorder characteriz | <br>ed by weakness and rapid fatigue of | any of the skeletal muscles. | | I | 1 |
| Neuralgia | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | _ | |
| veuraigia | Willia palli | instrumental ADL | ADL | - | - |
| Definition: A disorder characterize | ।<br>ed by intense painful sensation alona | 1 | 1 | 1 | , |
| Nystagmus | - | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| | | instrumental ADL | care ADL | | |
| Definition: A disorder characterize | ed by involuntary movements of the | eyeballs. | | | |
| Oculomotor nerve disorder | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| | diagnostic observations only; | instrumental ADL | care ADL | | |
| | intervention not indicated | | | | |
| Definition: A disorder characterize | ed by dysfunction of the oculomotor | nerve (third cranial nerve). | | | |
| Olfactory nerve disorder | - | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| | | instrumental ADL | care ADL | | |
| Definition: A disorder characterize | ed by dysfunction of the olfactory ne | erve (first cranial nerve). | T | T | |
| Paresthesia | Mild symptoms | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| | | instrumental ADL | care ADL | | |
| Definition: A disorder characterize | ed by functional disturbances of sens | sory neurons resulting in abnorma | cutaneous sensations of tingling, nu | mbness, pressure, cold, and/or v | varmth. |
| Peripheral motor neuropathy | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | Life-threatening | Death |
| | diagnostic observations only | instrumental ADL | care ADL | consequences; urgent | |
| | | | | intervention indicated | |
| Definition: A disorder characterize | ed by damage or dysfunctionof the p | peripheral motor nerves. | | T | |
| Peripheral sensory | Asymptomatic | Moderate symptoms; limiting | Severe symptoms; limiting self | Life-threatening | - |
| neuropathy | | instrumental ADL | care ADL | consequences; urgent | |
| Definition: A disorder characteriz | ed by damage or dysfunction of the | nerinheral sensory nerves | | intervention indicated | |
| Phantom pain | Mild pain | | Severe pain; limiting self care | _ | |
| -папсотт ратт | ivilia palii | Moderate pain; limiting<br>instrumental ADL | ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked discomf | T. | nat is removed from or is not physica | lly part of the body. | 1 |
| Presyncope | - | Present (eg, near fainting) | - | - | - |
| Definition: A disorder characteriz | ed by an episode of lightheadedness | and dizziness which may precede | an episode of syncope. | 1 | |
| Pyramidal tract syndrome | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | Life-threatening | Death |
| , | diagnostic observations only; | instrumental ADL | care ADL | consequences; urgent | |
| | intervention not indicated | | | intervention indicated | |
| | | | cord. Symptoms include an increase | in the muscle tone in the lower | extremiti |
| nyperreflexia, positive Babinski a | nd a decrease in fine motor coordina | ation. | | I | |
| Radiculitis | Mild symptoms | Moderate symptoms; medical | Severe symptoms; limiting self | Life-threatening | Death |
| | | intervention indicated; limiting | care ADL | consequences; urgent | |
| | | instrumental ADL | | intervention indicated | |

| | Grade | | | | |
|---|---|---|---|---|---|
| CTCAE Term | 1 | 2 | 3 | 4 | 5 |
| | Assumation district | | | life theretes in a | |
| Recurrent laryngeal nerve | Asymptomatic; clinical or | Moderate symptoms | Severe symptoms; medical | Life-threatening | Death |
| palsy | diagnostic observations only; | | intervention indicated | consequences; urgent | |
| | intervention not indicated | | (eg, thyroplasty, vocal cord | intervention indicated | |
| Definition: A disorder characterize | led by paralysis of the recurrent laryr | ogoal norvo | injection) | | l |
| | d by paralysis of the recurrent lary | | | | 5 |
| Reversible posterior | - | Moderate symptoms; | Severe symptoms; limiting | Life-threatening | Death |
| leukoencephalopathy | | limiting instrumental ADL | self care ADL; | consequences | |
| syndrome | Ţ | | hospitalization | | l |
| | ed by headaches, mental status cha | <del>-</del> ' | = = | | |
| | with hypertensive encephalopathy,<br>e encephalopathy syndrome (PRES). | | e and cytotoxic drug treatment. It is | an acute or subacute reversible cor | idition. |
| | | | Now onset sainures | Life threatening | Dooth |
| Seizure | Brief partial seizure and no loss | Brief generalized seizure | New onset seizures | Life-threatening | Death |
| | of consciousness | | (partial or generalized); | consequences; prolonged | |
| | | | multiple seizures despite | repetitive seizures | |
| | | | medical intervention | | l |
| Definition: A disorder characterize | ed by a sudden, involuntary skeletal | muscular contractions of cerebral of | r brain stem origin. | T | 1 |
| Somnolence | Mild but more than usual | Moderate sedation; limiting | Obtundation or stupor | Life-threatening | Death |
| | drowsiness or sleepiness | instrumental ADL | | consequences; urgent | |
| | | | | intervention indicated | |
| Definition: A disorder characterize | ed by excessive sleepiness and drow | siness. | | | |
| Spasticity | Mild or slight increase in | Moderate increase in muscle | Severe increase in muscle | Life-threatening consequences; | Death |
| | muscle tone | tone and increase in resistance | tone and increase in | unable to move active or | |
| | | through range of motion | resistance through range of | passive range of motion | |
| | | | motion | | |
| Definition: A disorder characteriz | ed by increased involuntary muscle | tone that affects the regions inte | rfering with voluntary movement. | It results in gait, movement, and s | peech |
| disturbances. | | | | | |
| Spinal cord compression | - | - | Severe symptoms; limiting self | Life-threatening | Death |
| | | | care ADL | consequences; urgent | |
| | | | | intervention indicated | |
| Definition: A disorder characterize | ed by pressure on the spinal cord. | | | | |
| | | | | | 1 |
| Stroke | Incidental radiographic | Mild to moderate | Severe neurologic deficit; | Life-threatening | Death |
| | findings only | neurologic deficit; limiting | limiting self care ADL; | consequences; urgent | |
| | | instrumental ADL | hospitalization | intervention indicated | |
| Definition: A disorder characterize | ed by a decrease or absence of blood | d supply to the brain caused by obst | ruction (thrombosis or embolism) o | f an artery resulting in neurological | damage |
| Syncope | - | - | Fainting; orthostatic collapse | - | - |
| Definition: A disorder characterize | ed by spontaneous loss of conscious | ness caused by insufficient blood su | pply to the brain. | | |
| Tendon reflux decreased | Ankle reflex reduced | Ankle reflex absent; other | Absence of all reflexes | - | - |
| | | reflexes reduced | | | |
| Definition: A disorder characteriz | ed by less than normal deep tendor | reflexes. | | | |
| Transient ischemic attacks | Mild noural agic doft-it!th | Moderate neurologic deficit | - | - | - |
| | Mild neurologic deficit with or | | | | |
| | Mild neurologic deficit with or without imaging confirmation | with or without imaging | | | |
| | without imaging confirmation | confirmation | | | |
| Definition: A disorder characterize | | confirmation | lar origin, with no persistent neurol | ogical deficit. | |
| | without imaging confirmation | confirmation | lar origin, with no persistent neurol<br>Severe symptoms; limiting self | ogical deficit. | - |
| | without imaging confirmation<br>ed by a brief attack (less than 24 hou | confirmation urs) of cerebral dysfunction of vascu | | ogical deficit. | - |
| Tremor | without imaging confirmation<br>ed by a brief attack (less than 24 hou | confirmation urs) of cerebral dysfunction of vascu Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | ogical deficit. | - |
| Tremor<br>Definition: A disorder characterize | without imaging confirmation ed by a brief attack (less than 24 hou Mild symptoms | confirmation urs) of cerebral dysfunction of vascu Moderate symptoms; limiting instrumental ADL ement of the whole body or individual. | Severe symptoms; limiting self care ADL lal parts. | ogical deficit. | - |
| Tremor<br>Definition: A disorder characterize | without imaging confirmation ed by a brief attack (less than 24 hou Mild symptoms ed by the uncontrolled shaking move Asymptomatic; clinical or | confirmation urs) of cerebral dysfunction of vascu Moderate symptoms; limiting instrumental ADL ement of the whole body or individu Moderate symptoms; limiting | Severe symptoms; limiting self care ADL lal parts. Severe symptoms; limiting self | ogical deficit. | - |
| Tremor<br>Definition: A disorder characterize | without imaging confirmation ed by a brief attack (less than 24 hou Mild symptoms ed by the uncontrolled shaking move | confirmation urs) of cerebral dysfunction of vascu Moderate symptoms; limiting instrumental ADL ement of the whole body or individual. | Severe symptoms; limiting self care ADL lal parts. | ogical deficit. | - |
| Tremor<br>Definition: A disorder characterize<br>Trigeminal nerve disorder | without imaging confirmation ed by a brief attack (less than 24 hou Mild symptoms ed by the uncontrolled shaking move Asymptomatic; clinical or diagnostic observations only; | confirmation urs) of cerebral dysfunction of vascu Moderate symptoms; limiting instrumental ADL ement of the whole body or individual Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL lal parts. Severe symptoms; limiting self | ogical deficit. | - |
| Tremor Definition: A disorder characterize Trigeminal nerve disorder Definition: A disorder characterize | without imaging confirmation ed by a brief attack (less than 24 hou Mild symptoms ed by the uncontrolled shaking move Asymptomatic; clinical or diagnostic observations only; intervention not indicated ed by dysfunction of the trigeminal red | confirmation urs) of cerebral dysfunction of vascu Moderate symptoms; limiting instrumental ADL mement of the whole body or individual instrumental ADL mereve (fifth cranial nerve). | Severe symptoms; limiting self care ADL ial parts. Severe symptoms; limiting self care ADL | ogical deficit. | - |
| Tremor<br>Definition: A disorder characterize<br>Trigeminal nerve disorder | without imaging confirmation ed by a brief attack (less than 24 hou Mild symptoms ed by the uncontrolled shaking move Asymptomatic; clinical or diagnostic observations only; intervention not indicated | confirmation urs) of cerebral dysfunction of vascu Moderate symptoms; limiting instrumental ADL ement of the whole body or individual Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL lal parts. Severe symptoms; limiting self | ogical deficit. - | - |

| Nervous system disord | lers | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| CTCAE Term | 1 | 2 | 3 | 4 | 5 |
| Vagus nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by dysfunction of the vagus nerve | (tenth cranial nerve). | | | |
| Vasovagal reaction | -<br>ed by a sudden drop of the blood pr | | Present | Life-threatening consequences; urgent intervention indicated | Death |
| the stimulation of the vagus nerve | | essure, bradycardia, and peripheral | vasoullation that may lead to loss t | or consciousness. It results from all | ilicrease ili |
| Nervous system disorders -<br>Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting<br>age-appropriate instrumental<br>ADL | Severe or medically significant<br>but not immediately<br>life-threatening; hospitalization<br>or prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

Abbreviations: ADL = activities of daily living; CTCAE = Common Terminology Criteria for Adverse Events; FLAIR = fluid-attenuated inversion recovery; ICP = intracranial pressure; PRES = posterior reversible encephalopathy syndrome; SAS = subarachnoid space.

| | Grade | | | | |
|---|---|---|---|---|---|
| CTCAE Term | | 2 | 3 | 4 | 5 |
| Agitation | Mild mood alteration | Moderate mood alteration | Severe agitation;<br>hospitalization not indicated | Life-threatening consequences; urgent intervention indicated | - |
| Definition: A disorder charac | terized by a state of restlessness associa | ।<br>ted with unpleasant feelings of irri | tability and tension. | I. | ı |
| Anorgasmia | Inability to achieve orgasm not adversely affecting relationship | Inability to achieve orgasm adversely affecting relationship | - | - | - |
| Definition: A disorder charac | terized by an inability to achieve orgasm | ·<br>I. | • | ' | " |
| Anxiety Definition: A disorder characteristics. | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL dread accompanied by restlessne | Severe symptoms; limiting self care ADL; hospitalization indicated | Life-threatening consequences; urgent intervention indicated ea unattached to a clearly identi | -<br>fiable |
| stimulus. | , | . , | | • | |
| Confusion | Mild disorientation | Moderate disorientation;<br>limiting instrumental ADL | Severe disorientation; limiting self care ADL | Life-threatening consequences; urgent | - |
| | | | | intervention indicated | |
| Definition: A disorder charac | terized by a lack of clear and orderly tho | | | intervention indicated | |
| Definition: A disorder charac<br>Delayed orgasm | terized by a lack of clear and orderly tho Delay in achieving orgasm not adversely affecting relationship | ught and behavior. Delay in achieving orgasm adversely affecting relationship | - | intervention indicated | - |
| Delayed orgasm | Delay in achieving orgasm not | Delay in achieving orgasm<br>adversely affecting<br>relationship | - | intervention indicated | - |
| Delayed orgasm | Delay in achieving orgasm not adversely affecting relationship | Delay in achieving orgasm<br>adversely affecting<br>relationship | Severe and acute confusional state; limiting self care ADL; urgent intervention indicated; new onset | Life-threatening consequences, threats of harm to self or others; urgent indicated | - Death |
| Delayed orgasm Definition: A disorder charace Delirium | Delay in achieving orgasm not<br>adversely affecting relationship<br>terized by sexual dysfunction characteriz | Delay in achieving orgasm adversely affecting relationship eed by a delay in climax. Moderate and acute confusional state; limiting instrumental ADL | state; limiting self care ADL;<br>urgent intervention indicated;<br>new onset | Life-threatening consequences, threats of harm to self or others; urgent intervention indicated | |

| | Grade | | | | |
|---|---|---|---|---|---|
| CTCAE Term | 1 | 2 | 3 | 4 | 5 |
| Depression | Mild depressive symptoms | Moderate depressive<br>symptoms; limiting<br>instrumental ADL | Severe depressive symptoms;<br>limiting self care ADL;<br>hospitalization not indicated | Life-threatening<br>consequences, threats of<br>harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characteri | zed by melancholic feelings of grief o | r unhappiness. | | | |
| Euphoria | Mild mood elevation | Moderate mood elevation | Severe mood elevation (eg, hypomania) | - | - |
| Definition: A disorder characteri | zed by an exaggerated feeling of wel | l-being which is disproportionate to | events and stimuli. | | |
| Hallucinations | Mild hallucinations (eg, perceptual distortions) | Moderate hallucinations | Severe hallucinations;<br>hospitalization not indicated | Life-threatening consequences, threats of harm to self or others; hospitalization indicated | Death |
| Definition: A disorder characteri | zed by a false sensory perception in | the absence of an external stimulus | | | _ |
| Insomnia | Mild difficulty falling asleep,<br>staying asleep or waking up<br>early<br>zed by difficulty in falling asleep and, | Moderate difficulty falling asleep, staying asleep or waking up early | Severe difficulty in falling asleep, staying asleep or waking up early | - | - |
| | | | | | T |
| Irritability | Mild/ easily consolable | Moderate; limiting instrumental ADL; increased attention indicated | Severe abnormal or excessive response; limiting self care ADL; inconsolable; medical or psychiatric intervention indicated | | - |
| Definition: A disorder character | ized by an abnormal responsiveness t | to stimuli or physiological arousal; m | nay be in response to pain, fright, a c | rug, an emotional situation or a mo | edical condi |
| Libido decreased | Decrease in sexual interest<br>not adversely affecting<br>relationship | Decrease in sexual interest adversely affecting relationship | - | - | - |
| Definition: A disorder characteri | zed by a decrease in sexual desire. | | | | |
| Libido increased | Present | - | - | - | - |
| Definition: A disorder characteri | zed by an increase in sexual desire. | ' | ' | • | |
| Mania | Mild manic symptoms (eg,<br>elevated mood, rapid<br>thoughts, rapid speech,<br>decreased need for sleep) | Moderate manic symptoms (eg, relationship and work difficulties; poor hygiene) | Severe manic symptoms (eg, hypomania; major sexual or financial indiscretions); hospitalization not indicated; | Life-threatening<br>consequences, threats of<br>harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characteri | zed by excitement of psychotic propo | ortions manifested by mental and p | hysical hyperactivity, disorganization | on of behavior and elevation of mo | od. |
| Personality change | Mild personality change | Moderate personality change | Severe personality change;<br>hospitalization not indicated | Life-threatening consequences, threats of harm to self or others; hospitalization indicated | - |
| Definition: A disorder characteri | zed by a conspicuous change in a per | rson's behavior and thinking. | T | | |
| Psychosis | Mild psychotic symptoms | Moderate psychotic symptoms<br>(eg, disorganized speech;<br>impaired reality testing) | Severe psychotic symptoms<br>(eg, paranoid; extreme<br>disorganization);<br>hospitalization not indicated;<br>new onset | Life-threatening<br>consequences, threats of<br>harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characteri | zed by personality change, impaired | functioning, and loss of touch with | reality. It may be a manifestation o | f schizophrenia, bipolar disorder o | r brain tum |
| Restlessness | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| | zed by an inability to rest, relax or be | | | | T |
| Suicidal ideation | Increased thoughts of death but no wish to kill oneself | Suicidal ideation with no specific plan or intent | Specific plan to commit suicide<br>without serious intent to die<br>which may not require | Specific plan to commit suicide<br>with serious intent to die<br>which requires hospitalization | - |

| Psychiatric disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| CTCAE Term | 1 | 2 | 3 | 4 | 5 |
| Suicide attempt | - | - | Suicide attempt or gesture without intent to die | Suicide attempt with intent to die which requires hospitalization | Death |
| Definition: A disorder characterize | ed by self-inflicted harm in an attem | npt to end one's own life. | | | |
| Psychiatric disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age- | · · | Life-threatening consequences;<br>hospitalization or urgent<br>intervention indicated | Death |
| | not indicated | appropriate instrumental ADL | self care ADL | | |

Abbreviations: ADL = activities of daily living; CTCAE = Common Terminology Criteria for Adverse Events.

# APPENDIX 3. ASBMT CONSENSUS GRADING SYSTEM OF IMMUNE EFFECTOR CELL-ASSOCIATED NEUROTOXICITY SYNDROME (ICANS) FOR ADULTS

| Neurotoxicity | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| ICE score <sup>a</sup> | 7-9 | 3-6 | 0-2 | 0 (patient is unarousable and unable to perform ICE) |
| Depressed level of consciousness <sup>b</sup> | Awakens<br>spontaneously | Awakens to voice | Awakens only to tactile stimulus | Patient is<br>unarousable or<br>requires vigorous or<br>repetitive tactile<br>stimuli to arouse.<br>Stupor or coma |
| Seizure | Not applicable | Not applicable | Any clinical seizure, focal or generalized that resolves rapidly; or nonconvulsive seizures on electroencephalogram that resolve with intervention | Life-threatening prolonged seizure (> 5 minutes); or repetitive clinical or electrical seizures without return to baseline in between |
| Motor findings <sup>c</sup> | Not applicable | Not applicable | Not applicable | Deep focal motor<br>weakness such as<br>hemiparesis or<br>paraparesis |
| Raised intracranial pressure/cerebral edema | Not applicable | Not applicable | Focal/local edema on neuroimaging <sup>d</sup> | Diffuse cerebral edema on neuroimaging; decerebrate or decorticate posturing; or cranial nerve VI palsy; or papilledema or Cushing's triad |

Note: ICANS grade is determined by the most severe event not attributable to any other cause. For example, a patient with an ICE score of 3 who has a generalized seizure is classified as having Grade 3 ICANS.

Abbreviations: CTCAE = Common Terminology Criteria for Adverse Events; ICANS = immune effector cell-associated neurotoxicity syndrome; ICE = immune effector cell-associated encephalopathy.

Source: Lee et al. 2019

<sup>&</sup>lt;sup>a</sup> A patient with an ICE score of 0 may be classified as Grade 3 ICANS if awake with global aphasia, but a patient with an ICE score of 0 may be classified as Grade 4 ICANS if unarousable.

<sup>&</sup>lt;sup>b</sup> Depressed level of consciousness should be attributable to no other cause (eg, no sedating medication).

<sup>&</sup>lt;sup>c</sup> Tremors and myoclonus associated with immune effector cell therapies may be graded according to CTCAE v5.0, but they do not influence ICANS grading.

<sup>&</sup>lt;sup>d</sup> Intracranial hemorrhage with or without associated edema is not considered a neurotoxicity feature and is excluded from ICANS grading. It may be graded according to CTCAE v5.0.

#### APPENDIX 4. GRADING OF CRS BY ASBMT CRITERIA

| CRS Parameter | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Fever <sup>a</sup> | Temperature ≥ 38°C | Temperature ≥ 38°C | Temperature ≥ 38°C | Temperature ≥ 38°C |
| With either: | | | | |
| Hypotension And/or <sup>b</sup> | None | Not requiring vasopressors | Requiring one vasopressor with or without vasopression | Requiring multiple<br>vasopressors<br>(excluding<br>vasopressin) |
| Hypoxia | None | Requiring low-flow<br>nasal cannula <sup>c</sup> or<br>blow-by | Requiring high-flow<br>nasal cannula <sup>c</sup> ,<br>facemask,<br>nonrebreather mask,<br>or Venturi mask | Requiring positive<br>pressure (eg, CPAP,<br>BiPAP, intubation<br>and mechanical<br>ventilation) |

Note: Organ toxicities associated with CRS may be graded according to CTCAE v5.0, but they do not influence CRS grading.

Source: Lee et al. 2019

<sup>&</sup>lt;sup>a</sup> Fever is defined as temperature ≥ 38°C not attributable to any other cause. In patients who have CRS then receive antipyretics or anticytokine therapy, such as tocilizumab or steroids, fever is no longer required to grade subsequent CRS severity. In this case, CRS grading is driven by hypotension and/or hypoxia.

<sup>&</sup>lt;sup>b</sup> CRS grade is determined by the more severe event: hypotension or hypoxia not attributable to any other cause. For example, a patient with termperature of 39.5°C, hypotension requiring 1 vasopressor, and hypoxia requiring low-flow nasal cannula is classified as having Grade 3 CRS.

c Low-flow nasal cannula is defined as oxygen delivered at ≤ 6 L/minute. Low flow also includes blow-by oxygen delivery, sometimes used in pediatrics. High-flow nasal cannula is defined as oxygen delivered at > 6 L/minute. Abbreviations: ASBMT = American Society of Blood and Marrow Transplant; BiPAP = bilevel positive airway pressure; CPAP = continuous positive airway pressure; CRS = cytokine release syndrome; CTCAE = Common Terminology Criteria for Adverse Events.

#### APPENDIX 5. MEDDRA 21.1 SMQ HAEMORRHAGE TERMS (EXCL LABORATORY TERMS)

Abdominal wall haematoma

Abdominal wall haemorrhage

Abnormal withdrawal bleeding

Achenbach syndrome

Acute haemorrhagic leukoencephalitis

Acute haemorrhagic ulcerative colitis

Administration site bruise

Administration site haematoma

Administration site haemorrhage

Adrenal haematoma

Adrenal haemorrhage

Anal fissure haemorrhage

Anal haemorrhage

Anal ulcer haemorrhage

Anastomotic haemorrhage

Anastomotic ulcer haemorrhage

Aneurysm ruptured

Angina bullosa haemorrhagica

Anorectal varices haemorrhage

Aortic aneurysm rupture

Aortic dissection rupture

Aortic intramural haematoma

Aortic perforation

Aortic rupture

Aponeurosis contusion

Application site bruise

Application site haematoma

Application site haemorrhage

Application site purpura

Arterial haemorrhage

Arterial intramural haematoma

Arterial perforation

Arterial rupture

Arteriovenous fistula site haematoma

Arteriovenous fistula site haemorrhage

Arteriovenous graft site haematoma

Arteriovenous graft site haemorrhage

Astringent therapy

Atrial rupture

Auricular haematoma

Basal ganglia haematoma

Basal ganglia haemorrhage

Basilar artery perforation

Bladder tamponade

Iris haemorrhage

Joint microhaemorrhage

Kidney contusion

Lacrimal haemorrhage

Large intestinal haemorrhage

Large intestinal ulcer haemorrhage

Laryngeal haematoma

Laryngeal haemorrhage

Lip haematoma

Lip haemorrhage

Liver contusion

Lower gastrointestinal haemorrhage

Lower limb artery perforation

Lymph node haemorrhage

Mallory-Weiss syndrome

Mediastinal haematoma

Mediastinal haemorrhage

Medical device site bruise

Medical device site haematoma

Medical device site haemorrhage

Melaena neonatal

Meningorrhagia

Menometrorrhagia

Menorrhagia

Mesenteric haematoma

Mesenteric haemorrhage

Metrorrhagia

Mouth haemorrhage

Mucocutaneous haemorrhage

Mucosal haemorrhage

Muscle contusion

Muscle haemorrhage

Myocardial haemorrhage

Myocardial rupture

Naevus haemorrhage

Nail bed bleeding

Nasal septum haematoma

Neonatal gastrointestinal haemorrhage

Nephritis haemorrhagic

Nipple exudate bloody

Ocular retrobulbar haemorrhage

Oesophageal haemorrhage

Oesophageal intramural haematoma

Bleeding varicose vein

Blood blister Blood urine

Blood urine present Bloody discharge

Bloody peritoneal effluent

Bone contusion

Bone marrow haemorrhage

Brain contusion

Brain stem haematoma Brain stem haemorrhage

Brain stem microhaemorrhage

Breast haematoma Breast haemorrhage

Broad ligament haematoma Bronchial haemorrhage

Bronchial varices haemorrhage

Bursal haematoma Cardiac contusion

Carotid aneurysm rupture Carotid artery perforation

Catheter site bruise

Catheter site haematoma Catheter site haemorrhage

Central nervous system haemorrhage

Cephalhaematoma
Cerebellar haematoma
Cerebellar haemorrhage
Cerebellar microhaemorrhage

Cerebral aneurysm perforation Cerebral aneurysm ruptured syphilitic

Cerebral arteriovenous malformation

haemorrhagic

Cerebral artery perforation

Cerebral haematoma Cerebral haemorrhage

Cerebral haemorrhage foetal Cerebral haemorrhage neonatal

Cerebral microhaemorrhage Cervix haematoma uterine

Cervix haemorrhage uterine

Chest wall haematoma Choroidal haematoma Choroidal haemorrhage

Chronic gastrointestinal bleeding

Chronic pigmented purpura

Oesophageal ulcer haemorrhage

Oesophageal varices haemorrhage

Oesophagitis haemorrhagic Optic disc haemorrhage

Optic nerve sheath haemorrhage

Oral contusion

Oral mucosa haematoma

Osteorrhagia

Ovarian haematoma
Ovarian haemorrhage
Palpable purpura

Pancreatic haemorrhage Pancreatitis haemorrhagic Papillary muscle haemorrhage Paranasal sinus haematoma Paranasal sinus haemorrhage

Parathyroid haemorrhage Parotid gland haemorrhage

Pelvic haematoma

Pelvic haematoma obstetric

Pelvic haemorrhage
Penile contusion
Penile haematoma
Penile haemorrhage
Peptic ulcer haemorrhage
Pericardial haemorrhage
Perineal haematoma
Periorbital haematoma
Periorbital haemorrhage
Periosteal haematoma

Peripartum haemorrhage

Peripheral artery aneurysm rupture Peripheral artery haematoma

Perirenal haematoma
Peritoneal haematoma
Peritoneal haemorrhage

Periventricular haemorrhage neonatal

Petechiae

Pharyngeal haematoma Pharyngeal haemorrhage Pituitary haemorrhage

Placenta praevia haemorrhage

Polymenorrhagia

Post abortion haemorrhage Post procedural contusion

Ciliary body haemorrhage

Coital bleeding
Colonic haematoma

Conjunctival haemorrhage

Contusion

Corneal bleeding

Cullen's sign

Cystitis haemorrhagic

Deep dissecting haematoma

Diarrhoea haemorrhagic

Disseminated intravascular coagulation

Diverticulitis intestinal haemorrhagic

Diverticulum intestinal haemorrhagic

Duodenal ulcer haemorrhage

Duodenitis haemorrhagic

Dysfunctional uterine bleeding

Ear haemorrhage

**Ecchymosis** 

Encephalitis haemorrhagic

Enterocolitis haemorrhagic

Epidural haemorrhage

**Epistaxis** 

Exsanguination

Extra-axial haemorrhage

Extradural haematoma

Extravasation blood

Eye contusion

Eye haematoma

Eye haemorrhage

Eyelid bleeding

**Eyelid** contusion

Eyelid haematoma

Femoral artery perforation

Femoral vein perforation

Foetal-maternal haemorrhage

Fothergill sign positive

Gastric haemorrhage

Gastric ulcer haemorrhage

Gastric ulcer haemorrhage, obstructive

Gastric varices haemorrhage

Gastritis alcoholic haemorrhagic

Gastritis haemorrhagic

Gastroduodenal haemorrhage

Gastrointestinal haemorrhage

Gastrointestinal polyp haemorrhage

Post procedural haematoma

Post procedural haematuria

Post procedural haemorrhage

Post transfusion purpura

Postmenopausal haemorrhage

Postpartum haemorrhage

Post-traumatic punctate intraepidermal

haemorrhage

Premature separation of placenta

Procedural haemorrhage

Proctitis haemorrhagic

Prostatic haemorrhage

Pulmonary alveolar haemorrhage

Pulmonary contusion

Pulmonary haematoma

Pulmonary haemorrhage

Puncture site haemorrhage

Purpura

Purpura fulminans

Purpura neonatal

Purpura non-thrombocytopenic

Purpura senile

Putamen haemorrhage

Radiation associated haemorrhage

Rectal haemorrhage

Rectal ulcer haemorrhage

Renal artery perforation

Renal cyst haemorrhage

Renal haematoma

Renal haemorrhage

Respiratory tract haemorrhage

Respiratory tract haemorrhage neonatal

Retinal aneurysm rupture

Retinal haemorrhage

Retinopathy haemorrhagic

Retroperitoneal haematoma

Retroperitoneal haemorrhage

Retroplacental haematoma

Ruptured cerebral aneurysm

Scleral haemorrhage

Scrotal haematocoele

Scrotal haematoma

Shock haemorrhagic

Skin haemorrhage

Skin neoplasm bleeding

Skin ulcer haemorrhage

Gastrointestinal ulcer haemorrhage

Gastrointestinal vascular malformation

haemorrhagic Genital contusion Genital haemorrhage Gingival bleeding Graft haemorrhage Grey Turner's sign

Haemarthrosis
Haematemesis

Haematochezia Haematocoele

Haematoma

Haematoma evacuation Haematoma infection

Haematosalpinx Haematospermia

Haematotympanum

Haematuria

Haematuria traumatic

Haemobilia

Haemophilic arthropathy
Haemophilic pseudotumour

Haemoptysis Haemorrhage

Haemorrhage coronary artery

Haemorrhage foetal

Haemorrhage in pregnancy
Haemorrhage intracranial
Haemorrhage neonatal
Haemorrhage subcutaneous
Haemorrhage subepidermal
Haemorrhage urinary tract

Haemorrhagic adrenal infarction

Haemorrhagic anaemia

Haemorrhagic arteriovenous malformation

Haemorrhagic ascites Haemorrhagic breast cyst

Haemorrhagic cerebral infarction

Haemorrhagic cyst Haemorrhagic diathesis

Haemorrhagic disease of newborn

Haemorrhagic disorder

Haemorrhagic erosive gastritis Haemorrhagic hepatic cyst Haemorrhagic infarction Small intestinal haemorrhage

Small intestinal ulcer haemorrhage

Soft tissue haemorrhage
Spermatic cord haemorrhage
Spinal cord haematoma
Spinal cord haemorrhage

Spinal epidural haematoma Spinal epidural haemorrhage

Spinal subarachnoid haemorrhage

Spinal subdural haematoma Spinal subdural haemorrhage

Spleen contusion

Splenic artery perforation Splenic haematoma Splenic haemorrhage

Splenic varices haemorrhage

Splinter haemorrhages
Spontaneous haematoma
Spontaneous haemorrhage
Stoma site haemorrhage
Stomatitis haemorrhagic
Subarachnoid haematoma
Subarachnoid haemorrhage

Subarachnoid haemorrhage neonatal

Subchorionic haematoma Subchorionic haemorrhage Subclavian artery perforation Subclavian vein perforation Subcutaneous haematoma Subdural haematoma

Subdural haematoma evacuation

Subdural haemorrhage

Subdural haemorrhage neonatal

Subgaleal haematoma Subgaleal haemorrhage Subretinal haematoma

Superior vena cava perforation

Testicular haemorrhage Thalamus haemorrhage

Third stage postpartum haemorrhage

Thoracic haemorrhage
Thrombocytopenic purpura

Thrombotic thrombocytopenic purpura

Thyroid haemorrhage Tongue haematoma

Haemorrhagic necrotic pancreatitis

Haemorrhagic ovarian cyst

Haemorrhagic stroke

Haemorrhagic thyroid cyst

Haemorrhagic transformation stroke

Haemorrhagic tumour necrosis

Haemorrhagic urticaria

Haemorrhagic vasculitis

Haemorrhoidal haemorrhage

Haemostasis

Haemothorax

Henoch-Schonlein purpura

Hepatic haemangioma rupture

Hepatic haematoma

Hepatic haemorrhage

Hereditary haemorrhagic telangiectasia

Hyperfibrinolysis

Hyphaema

Iliac artery perforation

Iliac artery rupture

Iliac vein perforation

Immune thrombocytopenic purpura

Implant site bruising

Implant site haematoma

Implant site haemorrhage

Incision site haematoma

Incision site haemorrhage

Increased tendency to bruise

Induced abortion haemorrhage

Inferior vena cava perforation

Infusion site bruising

Infusion site haematoma

Infusion site haemorrhage

Injection site bruising

Injection site haematoma

Injection site haemorrhage

Instillation site bruise

Instillation site haematoma

Instillation site haemorrhage

Internal haemorrhage

Intestinal haematoma

Intestinal haemorrhage

Intestinal varices haemorrhage

Intra-abdominal haematoma

Intra-abdominal haemorrhage

Intracerebral haematoma evacuation

Tongue haemorrhage

Tonsillar haemorrhage

Tooth pulp haemorrhage

Tooth socket haemorrhage

Tracheal haemorrhage

Traumatic haematoma

Traumatic haemorrhage

Traumatic haemothorax

Traumatic intracranial haematoma

Traumatic intracranial haemorrhage

Tumour haemorrhage

Ulcer haemorrhage

Umbilical cord haemorrhage

Umbilical haematoma

Umbilical haemorrhage

Upper gastrointestinal haemorrhage

Ureteric haemorrhage

Urethral haemorrhage

Urinary bladder haemorrhage

Urogenital haemorrhage

Uterine haematoma

Uterine haemorrhage

Vaccination site bruising

Vaccination site haematoma

Vaccination site haemorrhage

Vaginal haematoma

Vaginal haemorrhage

Varicose vein ruptured

Vascular access site bruising

Vascular access site haematoma

Vascular access site haemorrhage

Vascular access site rupture

Vascular graft haemorrhage

Vascular pseudoaneurysm ruptured

Vascular purpura

Vascular rupture

Vein rupture

Venous haemorrhage

Venous perforation

Ventricle rupture

Vertebral artery perforation

Vessel puncture site bruise

Vessel puncture site haematoma

Vessel puncture site haemorrhage

Vitreous haematoma

Vitreous haemorrhage

| Intracranial haematoma | Vulval haematoma |
|---------------------------------------|-----------------------------|
| Intracranial tumour haemorrhage | Vulval haematoma evacuation |
| Intraocular haematoma | Vulval haemorrhage |
| Intrapartum haemorrhage | Withdrawal bleed |
| Intraventricular haemorrhage | Wound haematoma |
| Intraventricular haemorrhage neonatal | Wound haemorrhage |